

Botanix BTX.2018.001

Version: v1

Date: 24 MAY 2019

# STATISTICAL ANALYSIS PLAN

Protocol Number: BTX.2018.001

Study Title: A Randomized, Double-Blind, Vehicle-

Controlled Study to Evaluate the Safety and Efficacy of BTX 1503 in Patients with Moderate to Severe Acne Vulgaris

Development Phase of Study: 2

Sponsor: Botanix Pharmaceuticals Ltd.

Sponsor Contact: Stephane Levy

Statistical Analysis Plan based on Protocol Version: 2.4 (07JUN2018)

Statistical Analysis Plan Date: 24 MAY 2019

Statistical Analysis Plan Version: v1

NCT03573518



Botanix BTX.2018.001

Version: v1 Date: 24 MAY 2019

SAP Approval

Authored by:

SIGNATURE;

Laura Hatsis, M.S. Manager of Statistics QST Consultations, Ltd. DATE: 2914A42019

Reviewed by:

SIGNATURE:

Lori Davis, Ph.D.

Associate Director of Biostatistical Consulting QST Consultations, Ltd.

DATE: 29May 2019

Approved by:

SIGNATURE.

Stephane Levy

Chief Medical Officer

Botanix

DATE: MAY 29 2019

Revisions to the Statistical Analysis Plan described herein must be approved through a formal written amendment with the exception of minor editorial changes to tables, figures, or listing shells, and any necessary textual clarifications for programmers that do not affect the stated analysis variables, study endpoints, or statistical methods.




Date: 24 MAY 2019

# SAP Change History

| Version | | Date | Summary of Changes | Author |
|---------|---|-----------|--------------------|--------------|
| | 1 | ddmmmyyyy | Original document | Laura Hatsis |



Botanix BTX.2018.001 Version: v1 Date: 24 MAY 2019

# TABLE OF CONTENTS

| 1. | LIS | T OF A | BBREVIATIONS AND DEFINITIONS OF TERMS | 6 |
|---|---|---|---|---|
| 2. | INTRODUCTION | | | |
| 3. | STI | IDY OB | BJECTIVES | 8 |
| 4. | STUDY DESIGN | | | |
| | 4.1 | | l Study Design | |
| | | 4.1.1 | Schedule of Visits and Assessments | |
| | | 4.1.2 | Method of Assigning Subjects to Treatment Groups | |
| | | 4.1.3 | Blinding | 9 |
| <b>5.</b> | EFI | FICACY | AND SAFETY ENDPOINTS | 9 |
| | 5.1 | Efficac | y Endpoints | 9 |
| | | 5.1.1 | Primary Efficacy Endpoint | 9 |
| | | 5.1.2 | Secondary Efficacy Endpoints | 9 |
| | | 5.1.3 | Exploratory Efficacy Endpoints | 10 |
| | 5.2 | Safety | Endpoints | 10 |
| 6. | STA | ATISTIC | CAL AND ANALYTICAL PLANS | 11 |
| | 6.1 | Genera | l Methodology | 11 |
| | | 6.1.1 | Statistical Analysis | 11 |
| | | 6.1.2 | Baseline Definition | 11 |
| | | 6.1.3 | Visit Windowing | 12 |
| | | 6.1.4 | Adjustments for Covariates | 12 |
| | | 6.1.5 | Handling of Dropouts or Missing Data | 13 |
| | | 6.1.6 | Interim Analyses and Data Monitoring | 13 |
| | | 6.1.7 | Multicenter Studies. | 13 |
| | | 6.1.8 | Multiple Comparisons/Multiplicity | 13 |
| | | 6.1.9 | Use of an Efficacy Subset of Subjects | 13 |
| | | 6.1.10 | Active-Control Studies Intended to Show Equivalence | 14 |
| | | 6.1.11 | Examination of Subgroups | 14 |
| | | | 6.1.11.1 Examination of Responders | |
| | 6.2 Disposition of Subjects | | | |
| | 6.3 Protocol Deviations | | | |
| | 6.4 | Data Se | ets Analyzed | 16 |



# Statistical Analysis Plan Botanix BTX.2018.001

Version: v1 Date: 24 MAY 2019

| | | 6.4.1 | Randomiz | zed Population | 16 |
|---|---|---|---|---|---|
| | | 6.4.2 | Intent-to- | Treat (ITT) Population | 16 |
| | | 6.4.3 | Safety Pop | pulation | 16 |
| | | 6.4.4 | Per-Protoc | col (PP) Population | 16 |
| | 6.5 | Demog | raphic and | Other Baseline Characteristics | 17 |
| | 6.6 | Prior a | nd Concom | itant Medications | 17 |
| | 6.7 | Concor | nitant Antil | biotic Therapies | 17 |
| | 6.8 | Analys | is of Effica | cy | 18 |
| | | 6.8.1 | Primary E | Efficacy Analysis | 18 |
| | | 6.8.2 | Secondary | y Efficacy Analysis | 18 |
| | | | 6.8.2.1 | Lesion Counts | 18 |
| | | | 6.8.2.2 | Investigator Global Assessment | 18 |
| | | 6.8.3 | Explorato | ry Efficacy Analysis | 19 |
| | | | 6.8.3.1 | Lesion Counts | 19 |
| | | | 6.8.3.2 | Investigator Global Assessment | 19 |
| | | | 6.8.3.3 | Acne-QoL | 20 |
| | | | 6.8.3.4 | Patient Reported Outcome (PRO) | 20 |
| | 6.9 | Sensiti | vity Analys | es | 20 |
| | 6.10 | Safety | Evaluation. | | 21 |
| | | 6.10.1 | Extent of | Exposure | 21 |
| | | 6.10.2 | Adverse E | Events | 22 |
| | | | 6.10.2.1 | Drug Abuse and Liability Assessments | 22 |
| | | 6.10.3 | Clinical L | aboratory Evaluation | 23 |
| | | 6.10.4 | Other Obs | servations Related to Safety | 23 |
| | | | 6.10.4.1 | Cutaneous Tolerability Assessments | 23 |
| | | | 6.10.4.2 | Physical Examination | 23 |
| <b>7.</b> | DET | ERMI | NATION ( | OF SAMPLE SIZE | 23 |
| 8. | CHA | NGES | IN THE P | PLANNED ANALYSES | 23 |
| 9. | REF | EREN | CES | | 23 |
| 10. | IND | EX OF | PLANNEI | D TABLES | 25 |
| 11. | IND | EX OF | PLANNEI | D LISTINGS | 150 |



Botanix BTX.2018.001


Date: 24 MAY 2019

#### 1. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AE(s) adverse event(s)

ANCOVA analysis of covariance

ATC anatomical therapeutic chemical

AUS Australia

BP blood pressure
BPM beats per minute

cm centimeters

CRF(s) case report form(s)

eCRF(s) electronic case report form(s)
FDA Food and Drug Administration

GCP good clinical practice

HEENT head, eyes, ears, nose, and throat

HR heart rate hr(s) hour(s)

ICH International Conference on Harmonization

ITT intent-to-treat kg kilograms

LOCF last observation carried forward

LSMean or LSM least squares mean

max maximum

MedDRA Medical Dictionary for Regulatory Activities

mg milligram min minimum

n number of observations

N number of subjects (sample size)

PP per-protocol PT preferred term

QST QST Consultations, Ltd. SAE(s) serious adverse event(s)

SAS® Statistical Analysis System (SAS® Institute Inc., Cary, NC)

SD standard deviation SOC system organ class



Botanix BTX.2018.001

Version: v1 Date: 24 MAY 2019

TEAE(s) treatment-emergent adverse event(s)

TEMP temperature
US United States

WHO World Health Organization

WHO-DDE World Health Organization Drug Dictionary

#### 2. INTRODUCTION

Acne is the most common skin disease in the world and is characterized by partial obstruction of the pores and associated local skin lesions that can appear on the face, chest or back [1, 2]. Obstructed pores can become enlarged and inflamed as sebum and its breakdown products accumulate, resulting in visible lesions that can be unsightly and cause permanent scarring [1, 2]. Acne usually begins in puberty and affects many adolescents and young adults, but it can occur at any stage of life. Approximately 85 percent of people between the ages of 12 and 24 experience at least minor acne [3]. Acne often causes significant physical and psychological problems such as permanent scarring, poor self-image, depression and anxiety [4].

Botanix Pharmaceuticals' BTX 1503 containing the active pharmaceutical ingredient, cannabidiol (CBD) in a topical liquid formulation, is being developed for the treatment of acne vulgaris. CBD is a member of a broader family of compounds knowns as cannabinoids, a class of compounds originally derived from the *cannabis sativa* plant [5].

No known well-controlled, human clinical studies have ever been conducted using CBD to treat skin disease, and no CDB containing pharmaceuticals have been approved to treat skin disease. Researchers have found that CBD may play a beneficial role in regulating the cutaneous endocannabinoid system by decreasing unwanted skin cell growth, sebum production and skin inflammation associated with many human skin diseases [5].

BTX 1503 is a formulation of active synthetic CBD and inactive excipients designed to deliver a consistent dose of CBD to directly treat patients with acne. It is considered that CBD may:

- normalize excessive lipid synthesis of human sebocytes;
- decrease proliferation (but not the viability) of these human sebocytes;
- inhibit hyperproliferation of keratinocytes;
- exert anti-inflammatory actions; and
- have anti-bacterial effects [5, 6].




This study is designed to investigate the efficacy, safety and tolerability of BTX 1503 in subjects with moderate to severe acne.

### 3. STUDY OBJECTIVES

The objective of this study is to assess safety and efficacy of various doses of BTX 1503 liquid formulation in subjects with moderate to severe acne vulgaris of the face.

#### 4. STUDY DESIGN

#### 4.1 Overall Study Design

This will be a multi-center, randomized, double-blind, vehicle-controlled, parallel group, dose-finding study in pediatrics, adolescents, and adults (aged 12 to 40 years). Approximately 360 subjects will be enrolled.

There will be five dose groups. All subjects will apply study drug for 84 days.

- BTX 1503 5% twice daily (BID),
- BTX 1503 5% once daily (QD),
- BTX 1503 2.5% once daily (QD),
- Vehicle BID, or
- Vehicle OD.

At the Baseline visit, qualified subjects will be randomized to treatment using an Interactive Web-based Randomization System (IWRS). The study will be a total of up to 17 weeks in duration; screening period up to 35 days (5 weeks) and 84 days (12 weeks) of treatment. During the study subjects will return to the study clinic at Day 14, 28, 56, and 84 (Study Exit).

#### 4.1.1 Schedule of Visits and Assessments

The schedule of assessments can be found in Section 7.3.8 of the protocol.

#### 4.1.2 Method of Assigning Subjects to Treatment Groups

A randomization schedule will be generated by a member in the QST Consultations, Ltd. (QST) Statistical Services department who is not associated with the conduct or analysis of the study, using a validated system. The randomization list will not be stratified, but stratification by site will be accomplished within the Interactive Web-based Randomization System (IWRS).




Once a subject is deemed eligible to enroll, randomization will occur using an IWRS. The IWRS will assign a study drug kit number based on a predetermined randomization schedule. The kit number will be recorded in the electronic case report form (eCRF). Randomization will be 2:2:2:1:1 (90 subjects in each active group and 45 in each vehicle group) and done by site.

#### 4.1.3 Blinding

The Sponsor, the CRO, the investigator, study site personnel and subjects will be blinded to the treatment assignment. The randomization schedule will be kept strictly confidential and accessible only to authorized persons. Only when the study has been completed, the protocol violations determined, and the study database locked will the randomization schedule be made available for analysis.

During the study, the randomization code will not be broken except in the case of a safety concern, either for an individual subject or for the entire study. If a subject has an adverse event (AE) that may necessitate unblinding of the randomization code, the site will contact the CRO and sponsor to discuss if there are options other than unblinding. If the site and sponsor agree that unblinding is in the best interests of the subject, the IWRS system will be used to obtain treatment assignment information. The Medical Monitor must be notified whenever study medication is unblinded, preferably prior to unblinding a subject.

#### 5. EFFICACY AND SAFETY ENDPOINTS

#### 5.1 Efficacy Endpoints

For all efficacy evaluations the measurement endpoint is defined at Day 84.

#### 5.1.1 Primary Efficacy Endpoint

The primary efficacy endpoint for the study is:

• Absolute change from Baseline in inflammatory lesion counts at Day 84.

#### **5.1.2** Secondary Efficacy Endpoints

The secondary efficacy endpoints for the study are:

- Absolute change from Baseline in non-inflammatory lesion counts at Day 84,
- The percent change from Baseline in the inflammatory lesion counts at Day 84,
- The percent change from Baseline in the non-inflammatory lesion counts at Day 84,




- The proportion of subjects with at least a 2-grade reduction from the Baseline IGA score at Day 84,
- The proportion of subjects with an IGA score of "clear" or "almost clear" at Day 84, and
- The proportion of subjects with an IGA score of "clear" or "almost clear" at Day 84 and at least a 2-grade reduction from the Baseline IGA score.

## **5.1.3** Exploratory Efficacy Endpoints

The exploratory efficacy endpoints are:

- The change from Baseline in the total lesion count at Day 84,
- The percent change from Baseline in the total lesion count at Day 84,
- The change from Baseline in the IGA scores at Day 84,
- The absolute and percent change from Baseline in inflammatory, non-inflammatory, and total lesion counts at Day 14, Day 28, and Day 56,
- The proportion of subjects with an IGA score of "clear" or "almost clear" at Day 14, Day 28, and Day 56,
- The proportion of subjects with at least a 2-grade reduction from the Baseline IGA score at Day 14, Day 28, and Day 56,
- The proportion of subjects with an IGA score of "clear" or "almost clear" at Day 14, Day 28, and Day 56 and at least a 2-grade reduction from the Baseline IGA score,
- The change from Baseline in the Acne-QoL at Day 84, and
- Subject's assessment of the change in their acne from Baseline to Day 84 (Patient Reported Outcome [PRO]).

### 5.2 Safety Endpoints

Safety will be assessed through adverse events (AEs), cutaneous tolerability (erythema, scaling, dryness, pruritus, and burning/stinging), complete blood count (CBC), chemistry, and urinalysis laboratory testing, and physical exam.




#### 6. STATISTICAL AND ANALYTICAL PLANS

# 6.1 General Methodology

All statistical processing will be performed using SAS® 9.3 or higher. No interim analyses are planned. This Phase 2 study is designed to identify the response to two different dosing frequencies and two concentrations of BTX 1503. Statistical tests applied to the outcomes will be exploratory. No adjustments for Type I error will occur.

Descriptive statistics will be used to provide an overview of the efficacy and safety results. For categorical parameters, the number and percentage of subjects in each category will be presented. For continuous parameters, descriptive statistics will include n (number of subjects), mean, standard deviation (SD), median, minimum and maximum.

The primary method of handling missing efficacy data in the ITT analysis set will be based on last observation carried forward (LOCF). Repeated measures analyses will be used on the observed data as a sensitivity analysis on the primary endpoint and the first secondary endpoint.

The efficacy analysis performed on the ITT population is considered the primary analysis. The efficacy analysis performed on the per-protocol (PP) population is considered supportive analysis.

The number of subjects in each analysis set will be summarized. Reasons for study withdrawal during the study will be summarized using frequencies and percentages by treatment group.

Reported AEs, medical history terms, and prior and concomitant procedures and therapies will be classified on the basis of Medical Dictionary for Regulatory Activities (MedDRA) terminology. Prior and concomitant medications will be classified on the basis of World Health Organization Drug Dictionary (WHO-DDE) terminology.

# **6.1.1** Statistical Analysis

All analyses will be performed by QST using SAS® Version 9.3 or later. All summary tables and data listings will be prepared utilizing SAS® software.

The standard operating procedures (SOPs) of QST will be followed in the creation and quality control of all data displays and analyses.

#### **6.1.2** Baseline Definition

Baseline is defined as the last non-missing assessment prior to first application of study drug.




# 6.1.3 Visit Windowing

Data will be summarized based on nominal visit indications with the exception of data captured at early termination and unscheduled visits. Data from early termination and unscheduled visits will be summarized based on mapped visit values. The analysis windows for early termination and unscheduled visits are presented in the following table.

#### **Analysis Windows**

| Scheduled Visit | Target Study Day | Window (Days) |
|-----------------|------------------|---------------|
| Day 14 | 15 | 9 to 21 |
| Day 28 | 29 | 22 to 42 |
| Day 56 | 57 | 43 to 70 |
| Day 84 | 85 | 71 to 98 |

Data collected at early termination and unscheduled visits prior to study day 9 will not be analyzed, with the exception of those identified as baseline values. Data collected at early termination and unscheduled visits after study day 98 will not be included in analyses.

The definition for the study day included in each study window is defined as below:

Study Day on or after Day 1 = Visit Date - Day 1 Date + 1

If an assessment's mapped visit is a visit at which the subject has data from a scheduled visit present, or if no analyses are planned for the assessment at the mapped visit, the data collected at the early termination or unscheduled visit will not be included in analyses.

In the event of multiple values from unscheduled or early termination assessments within an analysis window, the value closest to the scheduled visit target study day will be used for analyses. If two values tie as closest to the time point (for example, one value is before and the other value is after the time point), then the later value will be selected.

Data collected at all visits will be included in the data listings with visit presented as reported by the site.

## 6.1.4 Adjustments for Covariates

Baseline lesion count will be a covariate for the efficacy endpoints for acne lesion counts. No other covariates are planned to be used in the analyses for this study.




# 6.1.5 Handling of Dropouts or Missing Data

All efforts will be made to minimize the occurrence of missing data. It is not expected that dropout rates will differ between groups. Therefore, the primary method of handling missing efficacy data in the ITT analysis set will be based on last observation carried forward (LOCF). Summary of efficacy and pharmacology variables for the PP subjects will be based on available data. No imputation will be done for non-efficacy related variables.

If a partial date is reported where the day is missing, then the day will be imputed as the first day of the month unless the month is the same month as the first application of study drug then the day will be that of first application with the month and year remaining the same. If a partial date is reported where the month is missing, then the month will be imputed to January unless the year is the same year as the first application of study drug then the month will be that of first application with the year remaining the same. If a partial date where both the day and month is missing, follow details as stated previously.

Missing AE start dates will be imputed using partial date imputation rules as previously described in this Section.

#### 6.1.6 Interim Analyses and Data Monitoring

No interim analysis or data monitoring is planned for this study.

#### **6.1.7** Multicenter Studies

This study will be conducted at multiple investigational sites in the United States and Australia with the intention of pooling the results for analysis.

# 6.1.8 Multiple Comparisons/Multiplicity

This Phase 2 study is designed to identify the response to two different concentrations and dosing frequencies of BTX 1503. Statistical tests applied to the outcomes will be exploratory for establishing the dose and sample size for Phase 3 studies. No adjustments for Type I error will occur.

#### 6.1.9 Use of an Efficacy Subset of Subjects

Subjects randomized to study drug who complete the Day 84 visit without noteworthy study protocol violations, including compliance with study drug application, Day 84 visit window, and completion of efficacy evaluations on Day 84 will form the PP Population. The noteworthy




protocol violations will be defined at the time of evaluability evaluation, the time between the database soft lock and hard lock before unblinding.

Excluding subjects who have noteworthy protocol violations will decrease the variability in treatment response and will allow for a better determination of dose-response relationship of BTX 1503.

#### 6.1.10 Active-Control Studies Intended to Show Equivalence

Not applicable to this study.

#### **6.1.11** Examination of Subgroups

Subset analyses will be conducted for the PP analysis set on the primary efficacy endpoint and for the secondary endpoints, absolute change from Baseline in non-inflammatory lesion counts at Day 84 and subjects with an IGA score of "clear" or "almost clear" at Day 84 and at least a 2-grade reduction from the Baseline IGA score. These analyses will be summarized using descriptive statistics. The specific subsets within the PP analysis set that will be evaluated include:

- Baseline inflammatory lesion count (< median vs ≥ median);
- Baseline non-inflammatory count (< median vs ≥ median);
- Baseline total lesion count (< median vs ≥ median and < 80th percentile vs ≥ 80th percentile);</li>
- Baseline IGA (3 (Moderate) vs 4 (Severe));
- Baseline Acne-QoL:
  - $\circ$  Self-Perception domain (< median vs  $\geq$  median),
  - o Role-Social domain ( $\leq$  median vs  $\geq$  median),
  - o Role-Emotional (< median vs  $\ge$  median), and
  - o Acne Symptoms (< median vs  $\ge$  median);
- PRO (Improved (includes responses of much better and slightly better) vs. Same (includes response of the same) vs Worsened (includes responses of slightly worse and much worse));
- Geographical region (US vs AUS);



Botanix BTX.2018.001 Version: v1

- Gender (Male vs Female);

  Date: 24 MAY 2019
- Ethnicity (Hispanic or Latino vs Non-Hispanic or Latino);
- Race (White vs Non-White); and
- Age (12 to <18 vs 18 to <30 vs 30 to 40).

### **6.1.11.1 Examination of Responders**

Responder analyses will be conducted for the primary efficacy endpoint and for the secondary endpoints, absolute change from Baseline in non-inflammatory lesion counts at Day 84 and subjects with an IGA score of "clear" or "almost clear" at Day 84 and at least a 2-grade reduction from the Baseline IGA score. Responders are defined as, 80th percentile showing absolute reduction in inflammatory lesions from Baseline. These analyses will be summarized using descriptive statistics. The specific subsets within the responder PP analysis set that will be evaluated include:

- Baseline inflammatory lesion count (< median vs  $\ge$  median);
- Baseline non-inflammatory count (< median vs ≥ median);
- Baseline total lesion count (< median vs ≥ median and < 80th percentile vs ≥ 80th percentile);
- Baseline IGA (3 (Moderate) vs 4 (Severe));
- Compliance (percent compliance  $\leq$  median vs  $\geq$  median)

#### 6.2 Disposition of Subjects

The number of subjects included in each analysis population (randomized, ITT, safety, PP) will be summarized by treatment group. The number of subjects completed and discontinued (including the reasons for discontinuation) will be summarized for each treatment group.

Subjects who are excluded from an analysis population will be summarized by the reasons for exclusion.

#### **6.3** Protocol Deviations

Protocol deviations will not be entered into the database. Deviations leading to exclusion from analysis populations will be identified and summarized.




# 6.4 Data Sets Analyzed

# 6.4.1 Randomized Population

All subjects who are randomized to study treatment will be included in the randomized population and will be analyzed according to the treatment group they were randomized. Listings will be presented for all randomized subjects.

#### 6.4.2 Intent-to-Treat (ITT) Population

All subjects in the randomized population will be included in the ITT population and analyzed according to the randomized treatment group. All efficacy analyses will be presented using the ITT population.

#### **6.4.3** Safety Population

All subjects in the ITT population, who have at least one confirmed dose of study drug, and have at least one post-Baseline assessment will be included in the safety population and analyzed according to the treatment group received. All safety analyses will be performed using the safety population.

#### 6.4.4 Per-Protocol (PP) Population

All subjects in the ITT population who complete the Day 84 visit without noteworthy study protocol violations will be included in the PP population and analyzed according to the treatment group received. The PP population will include subjects in the ITT population who do not meet any of the following criteria:

- Violated the inclusion/exclusion criteria;
- Have taken any interfering concomitant medication;
- Did not complete both IGA and lesion count efficacy assessments at the Day 84 visit;
- Have missed both the Day 28 and Day 56 visits;
- Have not been compliant with the dosing regimen (i.e. subjects must apply 80-120% of the expected applications of study medication during participation in the study);
- Out of visit window at the Day 84 visit by  $\pm 5$  days;

Subjects that discontinue from the study due to an AE related to study treatment or documented lack of treatment effect will be included in the PP population. Prior to breaking the blind, other




additional criteria may be added to the list to accommodate for unforeseen events that occurred during the conduct of the trial that result in noteworthy study protocol violations.

All efficacy analyses will be performed on the PP population.

#### 6.5 Demographic and Other Baseline Characteristics

All demographic and Baseline summaries will be done on the ITT, PP, and safety populations.

Sex, race, and ethnicity will be summarized by counts and percentages. Age, height (cm), and weight (kg) will be summarized with descriptive statistics.

Tobacco and alcohol history will be summarized with counts and percentages. Baseline IGA and inflammatory and non-inflammatory lesion counts will be summarized with descriptive statistics.

Medical histories will be coded using the MedDRA dictionary and presented in a by-subject listing.

#### 6.6 Prior and Concomitant Medications

Concomitant medications will be coded to preferred name and Anatomical Therapeutic Chemical (ATC) classification of ingredients using the World Health Organization (WHO) Drug dictionary (WHO-DDE).

Counts and percentages will be provided to summarize the use of concomitant medications other than the study drug reported throughout the study. The number and percent of subjects who took other therapy will be shown by ATC level 2 term and preferred name. Medications which start prior to first application will be considered prior medications. Ongoing medications and medications ending after the date of first application will be considered concomitant medications. Incomplete start and end dates which could be either prior to first application or after first application will be considered prior to first application.

A by-subject listing of all prior and concomitant medications will be presented.

#### 6.7 Concomitant Antibiotic Therapies

Concomitant antibiotic therapies will be determined by the sponsor prior to database lock.

Counts and percentages will be provided to summarize the use of concomitant antibiotic therapies reported throughout the study. The number and percent of subjects who took concomitant antibiotic therapies will be shown by ATC level 2 term and preferred name.

A by-subject listing of all concomitant antibiotic therapies will be presented.




# 6.8 Analysis of Efficacy

The efficacy analyses will be performed using the ITT (primary) and PP (supportive) analysis sets. The lesion count and IGA analyses will employ the methods for handling missing data as described by Section 6.1.5. Lesion count and IGA data will also be shown in by-subject listings.

#### 6.8.1 Primary Efficacy Analysis

Absolute change from Baseline to Day 84 in inflammatory lesion counts will be analyzed using either parametric or non-parametric methods consistent with the statistical assumptions required to support the analyses. Specifically, the tests of superiority will be based on an ANCOVA with factors of treatment (with the vehicle treatment groups combined) and the respective Baseline lesion count as a covariate, or on ranked data submitted to an ANCOVA with factors of treatment and the respective Baseline lesion count as a covariate.

A skewness test, based on the methods presented by J.H. Zar (1984), will be applied to the residuals resulting from an ANCOVA. A two-sided p-value for the skewness test significant at 0.01 will imply the use of the non-parametric method. If a parametric analysis is indicated, the results of the parametric analysis will be considered the primary analysis. Should a non-parametric analysis be indicated, the absolute changes in inflammatory lesions will be rank transformed prior to submitting them to the ANCOVA. Results of the rank-transformed analyses then will be considered the primary analysis; however, results of the non-ranked transformed analyses will also be presented.

#### 6.8.2 Secondary Efficacy Analysis

#### 6.8.2.1 Lesion Counts

The absolute change from Baseline in non-inflammatory lesion count at Day 84 will be summarized similarly as absolute change from Baseline for inflammatory lesion count (primary efficacy endpoint). Percent change from Baseline to Day 84 in inflammatory and non-inflammatory lesion counts will be analyzed using the same ANCOVA method described for the primary endpoint.

#### 6.8.2.2 Investigator Global Assessment

The proportion of subjects with at least a 2-grade reduction from the Baseline IGA score at Day 84 will be analyzed with logistic regression. Pairwise tests will be conducted comparing the treated groups to a combined vehicle. The proportion of subjects with an IGA score of "clear" or "almost clear" at Day 84 will be analyzed using the same logistic method as described above.




Date: 24 MAY 2019

The IGA will be dichotomized into "success" and "failure", with a subject considered a "success" at each individual visit if the IGA at that visit is Clear ("0") or Almost Clear ("1") and at least 2 grades less than the Baseline score. The proportion of subjects who are dichotomized to success at Day 84 will be analyzed using the same logistic method as described above.

#### **6.8.3** Exploratory Efficacy Analysis

#### 6.8.3.1 Lesion Counts

The absolute and percent change from Baseline in the total lesion count at Day 84 will be summarized with descriptive statistics.

Additional comparisons between vehicle BID to BTX 1503 BID and vehicle QD to each BTX 1503 QD group for the absolute and percent change from Baseline to Day 84 in inflammatory and non-inflammatory lesion counts will be analyzed using either parametric or non-parametric methods consistent with the approach used for the primary endpoint using an ANCOVA with factors of treatment where no treatment groups are combined and the respective Baseline lesion count as a covariate or on ranked data submitted to an ANCOVA with factors of treatment where no treatment groups are combined and the respective Baseline lesion count as a covariate.

A further comparison will be made between vehicle QD to a combined BTX 1503 QD group for the absolute and percent change from Baseline to Day 84 in inflammatory and non-inflammatory lesion counts using an ANCOVA with factors of treatment where the two BTX 1503 QD treatment groups are combined and the respective Baseline lesion count as a covariate or on ranked data submitted to an ANCOVA with factors of treatment where the two BTX 1503 QD treatment groups are combined and the respective Baseline lesion count as a covariate.

The absolute and percent change from Baseline in inflammatory, non-inflammatory, and total lesion counts will be summarized at Day 14, Day 28, and Day 56. The absolute and percent change from Baseline in inflammatory, non-inflammatory, and total lesion counts at Day 14, Day 28, and Day 56 will be analyzed using the same ANCOVA method used for the primary endpoint as well as the additional testing described above in this section.

#### 6.8.3.2 Investigator Global Assessment

The dichotomized IGA success at Day 84 will be analyzed with an additional logistic regression analysis where no treatment groups are combined. Pairwise tests will be conducted comparing the vehicle BID to BTX 1503 BID and comparing the vehicle QD to each BTX 1503 QD group. The dichotomized IGA success at Day 84 will additionally be analyzed with a logistic regression




where the two BTX 1503 QD treatment groups are combined. Pairwise tests will be conducted comparing the vehicle QD to BTX 1503 QD combined.

The change from Baseline in the IGA scores at Day 14, Day 28, Day 56, and Day 84 will be summarized with descriptive statistics. The proportion of subjects who are dichotomized to success at Day 14, Day 28, and Day 56 will be summarized with proportions. The dichotomized success at Day 14, Day 28, and Day 56 will also be analyzed using the same logistic method as in the secondary efficacy analysis as well as the additional testing described above in this section.

## 6.8.3.3 Acne-QoL

The change from Baseline in the Acne-QoL domain scores at Day 84 will be summarized with descriptive statistics by domain score and treatment group. Domains for the Acne-QoL include Self-Perception, Role-Social, Role-Emotional, and Acne Symptoms. Responses will be coded numerically on a scale from 0 ('extremely' or 'extensive') to 6 ('not at all' or 'none') within each domain. All questions in each domain will be summed to get the total domain score.

Self-Perception includes Q1, Q2, Q3, Q6, and Q10; Role-Social includes Q11, Q12, Q13, and Q14; Role-Emotional includes Q4, Q5, Q7, Q8, and Q9; and Acne Symptoms includes Q15, Q16, Q17, Q18, and Q19 (Martin 2001).

Domain scores as well as individual question responses will be listed in a by-subject listing.

#### 6.8.3.4 Patient Reported Outcome (PRO)

The PRO will be summarized with counts and percentages by treatment group.

PRO results will also be shown in a by-subject listing.

#### 6.9 Sensitivity Analyses

A sensitivity analysis will be performed using the ITT population. The primary and the first secondary endpoints (change from Baseline in inflammatory and non-inflammatory lesion counts) will be analyzed using a repeated measures ANCOVA, with treatment group and visit as independent factors and the Baseline value as a covariate.

```
proc mixed data = datain method = ML;
  class SUBJECT TRT VISIT;
  model CHG = TRT VISIT TRT * VISIT BASE / solution;
  repeated VISIT / subject = SUBJECT type = cs;
  lsmeans TRT | VISIT / diff;
run;
```




# 6.10 Safety Evaluation

# **6.10.1** Extent of Exposure

The extent of exposure to study drug in each treatment group will be summarized by total number of days of exposure, total number of applications, number of missed applications, number and percentage of subjects who are compliant, average amount of study drug used per day (g/day), and amount of drug used total (g). A subject will be considered compliant with the dosing regimen if the subject applied 80% to 120% of the expected number of applications while enrolled in the study.

The total amount of study drug used will be calculated from the drug accountability using the recorded weights. The difference between the dispensed weight and the returned weight for each pump will be summed over all pumps to get the total amount of study drug used. The total amount of study drug used will be divided by the total number of exposure days to get the average amount of study drug used per day.

The total number of days of exposure is as follows:

Date of Last Application – Date of First Application + 1.

It will be assumed the BID subjects were expected to have 2 applications on the Date of First Application. It will also be assumed the BID subjects were expected to have only 1 application on the Date of Last Application unless there is evidence to suggest otherwise (i.e. dosing deviation log indicates 2 doses were expected).

The total number of applications taken for BID subjects is as follows:

2 applications expected on Date of Last Application: 2\*(Date of Last Application – Date of First Application + 1) – (Number of doses marked as missed on the CRF);

1 application expected on Date of Last Application: 2\*(Date of Last Application – Date of First) + 1 – (Number of doses marked as missed on the CRF).

The total number of applications taken for QD subjects is as follows:

(Date of Last Application – Date of First Application + 1) – (Number of doses marked as missed on the CRF).

The total number of applications expected for BID subjects is as follows:

2 applications expected on Date of Last Application: 2\*(Date Subject Ended Participation

- Date of Randomization + 1);




Date: 24 MAY 2019

1 application expected on Date of Last Application: 2\*(Date Subject Ended Participation – Date of Randomization) + 1.

The total number of applications expected for QD subjects is as follows:

Date Subject Ended Participation – Date of Randomization + 1.

If the total number of applications for BID subjects exceeds 178 then it will be set to 178.

If the total number of applications for QD subjects exceeds 89 then it will be set to 89.

Compliance will be calculated as a percentage as 100 times the total number of applications taken divided by the total number of applications expected while enrolled in the study.

#### 6.10.2 Adverse Events

All AEs that occur during the study will be recorded and classified on the basis of Medical Dictionary for Regulatory Activities (MedDRA) terminology. Treatment-emergent AEs (TEAEs) are defined as AEs with an onset on or after the date of the first study drug application. Adverse events noted prior to the first study drug administration that worsen after Baseline will also be reported as AEs and included in the summaries.

An overall summary of TEAEs will be presented showing the number of subjects reporting at least one TEAE, number reporting at least one SAE, number reporting at least one TEAE leading to study discontinuation, and number of TEAEs by severity and by relationship for each treatment group. The total number of AEs will also be presented as part of the overall summary of TEAEs. Treatment-emergent AEs will be summarized by system organ class and preferred name. Serious TEAEs, Related TEAEs, Severe TEAEs, and TEAEs leading to study discontinuation will also be summarized by system organ class and preferred name.

In addition, a listing of all AEs, a listing of Serious AEs, and a listing of subjects who prematurely discontinue from the study due to an AE will be provided.

No statistical inference between treatments will be performed on AEs.

# 6.10.2.1 Drug Abuse and Liability Assessments

Adverse events associated with potential abuse or overdose will be recorded and classified by MedDRA System Organ Classifications (SOC) and MedDRA Preferred Terms (PTs) as outlined in the Safety Management Plan. The incidence of abuse related AEs will be summarized by treatment group using frequency counts and percentages.

A by-subject listing of abuse related AEs will also be presented.




# 6.10.3 Clinical Laboratory Evaluation

Laboratory test results will be summarized with descriptive statistics at Baseline and Day 84. Additionally, shifts from Baseline to Day 84 in laboratory test results based on normal ranges will be summarized with frequency counts and percentages. Individual laboratory test results as well as pregnancy test results will be presented in a by-subject listing.

### 6.10.4 Other Observations Related to Safety

#### **6.10.4.1 Cutaneous Tolerability Assessments**

Cutaneous tolerability (erythema, scaling, dryness, pruritus, and burning/stinging) will be summarized at each visit using counts and percentages by treatment group. In addition, worst post-Baseline grade will be summarized by treatment group using counts and percentages. Any incident of mild, moderate, or severe post-Baseline results will be summarized by treatment group using counts and percentages.

## 6.10.4.2 Physical Examination

Physical examination data will be presented in a by-subject listing.

#### 7. DETERMINATION OF SAMPLE SIZE

The sample size for this study is based on clinical considerations only. Subjects will be randomized 2:2:2:1:1 with 90 subjects in each active treatment group and 45 subjects in each vehicle group for a total 360 subjects. This is considered adequate to evaluate the safety and tolerability of BTX 1503 in the treatment of acne vulgaris.

#### 8. CHANGES IN THE PLANNED ANALYSES

There are no changes in the conduct of the study or planned analyses.

#### 9. REFERENCES

- 1. Katsambas A, Papakonstantinou A. Acne: system treatment. *Clinics in Dermatology* 2004;22:412-8
- 2. Bhate K, Williams HC. What's new in acne? An analysis of systematic reviews published in 2011-2012. *Clinical and Experimental Dermatology* 2014;39:273-7; quiz 7-8
- 3. Bhate K, Williams HC. Epidemiology of acne vulgaris. *The British Journal of Dermatology* 2013;168:474-85




- 4. Strauss JS, Krowchuk DP, Leyden JJ, Lucky AW, Shalita AR, Siegfried EC et al. Guidelines of care for acne vulgaris management. *Journal of the American Academy of Dermatology* 2007;56:651-6
- 5. Olah A, Toth B, Borbiro I, et al, Cannabidiol exerts sebostatic and anti-inflammatory effects on human sebocytes, J Clin Invest 2014; 124(9); 3713-3724
- 6. van Klingeren B, ten Ham M, Antibacterial activity of Δ9-tetrahydrocannabionol and cannabidiol *Antoine van Leeuwenhoek* 1976; 42: 9-12




Date: 24 MAY 2019

# 10. INDEX OF PLANNED TABLES

| Table 14.0.1: Summary of Subject Completion/Discontinuation (Randomized Subjects) | 30 |
|---|---|
| Table 14.0.2: Summary of Subjects Excluded from Analyses (Randomized Subjects) | 31 |
| Table 14.0.3: Summary of Reasons for Screen Failure (Non-Randomized Subjects) | 32 |
| Table 14.1.1.1: Summary of Subject Demographics (ITT Population) | 33 |
| Table 14.1.1.2: Summary of Subject Demographics (PP Population) | 35 |
| Table 14.1.1.3: Summary of Subject Demographics (Safety Population) | 35 |
| Table 14.1.2.1: Summary of Baseline Characteristics (ITT Population) | 36 |
| Table 14.1.2.2: Summary of Baseline Characteristics (PP Population) | 38 |
| Table 14.1.2.3: Summary of Baseline Characteristics (Safety Population) | 38 |
| Table 14.1.3.1: Summary of Concomitant Medications by ATC Level 2 Term and Preferred Name (ITT Population) | 39 |
| Table 14.1.3.2: Summary of Concomitant Medications by ATC Level 2 Term and Preferred Name (PP Population) | 40 |
| Table 14.1.3.3: Summary of Concomitant Medications by ATC Level 2 Term and Preferred Name (Safety Population) | 40 |
| Table 14.1.4.1: Summary of Concomitant Antibiotic Therapies by ATC Level 2 Term and Preferred Name (ITT Population) | 41 |
| Table 14.1.4.2: Summary of Concomitant Antibiotic Therapies by ATC Level 2 Term and Preferred Name (PP Population) | 42 |
| Table 14.1.4.3: Summary of Concomitant Antibiotic Therapies by ATC Level 2 Term and Preferred Name (Safety Population) | 42 |
| Table 14.2.1.1: Primary Efficacy Endpoint: Summary of Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (ITT Population) | 43 |
| Table 14.2.1.2: Primary Efficacy Endpoint: Summary of Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population) | 44 |
| Table 14.2.1.3: Sensitivity Analysis of Primary Efficacy Endpoint: Summary of Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (IT Population) | |
| Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline Inflammatory Lesion Count at Day 84 (PP Population) | |
| Table 14.2.1.4: Responder Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population - Responders) | |



| Statio | ctical | Ana | lveic | Dlan |
|--------|---------|-----|-------|------|
| SIBLE | 211('%1 | Апя | | PINI |

| Date: 24 MAY 2019 |
|---|
| Table 14.2.2.1.1: Secondary Efficacy Endpoint: Summary of Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (ITT Population)67 |
| Table 14.2.2.1.2: Secondary Efficacy Endpoint: Summary of Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population)68 |
| Table 14.2.2.1.3: Sensitivity Analysis of Secondary Efficacy Endpoint: Summary of Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (ITT Population) |
| Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) |
| Table 14.2.2.1.5: Responder Subgroup Summary of the Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population - Responders) |
| Table 14.2.2.2.1: Secondary Efficacy Endpoint: Summary of Percent Change from Baseline in Inflammatory and Non-Inflammatory Lesion Count at Day 84 (ITT Population) |
| Table 14.2.2.2: Secondary Efficacy Endpoint: Summary of Percent Change from Baseline in Inflammatory and Non-Inflammatory Lesion Count at Day 84 (PP Population) |
| Table 14.2.2.3.1: Secondary Efficacy Endpoint: Summary of Dichotomized IGA at Day 84 (ITT Population) |
| Table 14.2.2.3.2: Secondary Efficacy Endpoint: Summary of Dichotomized IGA at Day 84 (PP Population) |
| Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population)96 |
| Table 14.2.2.3.4: Responder Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population - Responders)110 |
| Table 14.2.3.1.1: Exploratory Efficacy Endpoint: Summary of Inflammatory Lesion Count by Visit (ITT Population) |
| Table 14.2.3.1.2: Exploratory Efficacy Endpoint: Summary of Inflammatory Lesion Count by Visit (PP Population) |
| Table 14.2.3.2.1: Exploratory Efficacy Endpoint: Summary of Non-Inflammatory Lesion Count by Visit (ITT Population) |
| Table 14.2.3.2.2: Exploratory Efficacy Endpoint: Summary of Non-Inflammatory Lesion Count by Visit (PP Population) |
| Table 14.2.3.3.1: Exploratory Efficacy Endpoint: Summary of Total Lesion Count by Visit (ITT Population) |




| | Date: 24 MAY 2019 fficacy Endpoint: Summary of Total Lesion Count by Visit opulation)117 |
|---|---|
| Baseli | fficacy Endpoint: Analysis of Absolute and Percent Change from ne in Inflammatory Lesion Count at Day 84 (Comparing Dose encies) (ITT Population) |
| Baseli | fficacy Endpoint: Analysis of Absolute and Percent Change from ne in Inflammatory Lesion Count at Day 84 (Comparing Dose encies) (PP Population) |
| Baseli | fficacy Endpoint: Analysis of Absolute and Percent Change from ne in Non-Inflammatory Lesion Count at Day 84 (Comparing Frequencies) (ITT Population) |
| Baseli | fficacy Endpoint: Analysis of Absolute and Percent Change from ne in Non-Inflammatory Lesion Count at Day 84 (Comparing Frequencies) (PP Population) |
| 1 | fficacy Endpoint: Analysis of Absolute and Percent Change from ne in Inflammatory Lesion Count by Visit (ITT Population)121 |
| | fficacy Endpoint: Analysis of Absolute and Percent Change from ne in Inflammatory Lesion Count by Visit (PP Population)123 |
| Baseli | fficacy Endpoint: Analysis of Absolute and Percent Change from ne in Non-Inflammatory Lesion Count by Visit Population) |
| Baseli | fficacy Endpoint: Analysis of Absolute and Percent Change from ne in Non-Inflammatory Lesion Count by Visit opulation) |
| 1 | fficacy Endpoint: Analysis of Absolute and Percent Change from ne in Total Lesion Count by Visit (ITT Population)123 |
| | fficacy Endpoint: Analysis of Absolute and Percent Change from ne in Total Lesion Count by Visit (PP Population)123 |
| Baseli | fficacy Endpoint: Analysis of Absolute and Percent Change from ne in Inflammatory Lesion Count by Visit (Comparing Dose encies) (ITT Population) |
| Baseli | fficacy Endpoint: Analysis of Absolute and Percent Change from ne in Inflammatory Lesion Count by Visit (Comparing Dose encies) (PP Population) |
| from I | Efficacy Endpoint: Analysis of Absolute and Percent Change Baseline in Non-Inflammatory Lesion Count by Visit (Comparing Frequencies) (ITT Population) |




| Date: 24 MAY | |
|---|---|
| Table 14.2.3.10.2: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Non-Inflammatory Lesion Count by Visit (Compa Dose Frequencies) (PP Population) | ring |
| Table 14.2.3.11.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Total Lesion Count by Visit (Comparing Dose Frequencies) (ITT Population) | |
| Table 14.2.3.11.2: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Total Lesion Count by Visit (Comparing Dose Frequencies) (PP Population) | |
| Table 14.2.3.12.1: Exploratory Efficacy Endpoint: Summary of IGA Score by Visit (ITT Population) | .131 |
| Table 14.2.3.12.2: Exploratory Efficacy Endpoint: Summary of IGA Score by Visit (PP Population) | .132 |
| Table 14.2.3.13.1: Exploratory Efficacy Endpoint: Analysis of Dichotomized IGA at Day 84 (Comparing Dose Frequencies) (ITT Population) | .133 |
| Table 14.2.3.13.2: Exploratory Efficacy Endpoint: Analysis of Dichotomized IGA at Day 84 (Comparing Dose Frequencies) (PP Population) | .134 |
| Table 14.2.3.14.1: Exploratory Efficacy Endpoint: Analysis of Dichotomized IGA by Visit (I Population) | |
| Table 14.2.3.14.2: Exploratory Efficacy Endpoint: Analysis of Dichotomized IGA by Visit (PP Population) | .136 |
| Table 14.2.3.15.1: Exploratory Efficacy Endpoint: Analysis of Dichotomized IGA by Visit (Comparing Dose Frequencies) (ITT Population) | .137 |
| Table 14.2.3.15.2: Exploratory Efficacy Endpoint: Analysis of Dichotomized IGA by Visit (Comparing Dose Frequencies) (PP Population) | .138 |
| Table 14.2.3.16.1: Exploratory Efficacy Endpoint: Summary of Acne Patient Self-Questionna (ITT Population) | |
| Table 14.2.3.16.2: Exploratory Efficacy Endpoint: Summary of Acne Patient Self-Questionna (PP Population) | aire |
| Table 14.2.3.17.1: Exploratory Efficacy Endpoint: Summary of Patient Reported Outcome (I' Population) | |
| Table 14.2.3.17.2: Exploratory Efficacy Endpoint: Summary of Patient Reported Outcome (PP Population) | .142 |
| Table 14.3.0.1: Summary of Extent of Exposure (Safety Population) | .143 |
| Table 14.3.0.2.1: Summary of Cutaneous Tolerability Assessments (Safety Population) | .145 |




| Table 14.3.0.2.2: Summary of Cutaneous Tolerability Assessments Worst Post-Baseline Grades (Safety Population) |
|---|
| Table 14.3.0.2.3: Summary of Mild, Moderate, or Severe Post-Baseline Cutaneous Tolerability Assessments (Safety Population) |
| Table 14.3.1.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population) |
| Table 14.3.1.1.2: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)149 |
| Table 14.3.1.1.3: Summary of Serious Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)150 |
| Table 14.3.1.1.4: Summary of Related Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)150 |
| Table 14.3.1.1.5: Summary of Severe Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)150 |
| Table 14.3.1.1.6: Summary of Treatment-Emergent Adverse Events Leading to Study Discontinuation by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.1.7: Summary of Treatment-Emergent Abuse-Related Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)150 |
| Table 14.3.1.2.1.1: Summary of Chemistry Results by Visit (Safety Population)151 |
| Table 14.3.1.2.1.2: Shift Table for Chemistry Results (Safety Population) |
| Table 14.3.1.2.2.1: Summary of CBC Results by Visit (Safety Population) |
| Table 14.3.1.2.2.2: Shift Table for CBC Results (Safety Population) |
| Table 14.3.1.2.3.1: Summary of Numeric Urinalysis Results by Visit (Safety Population)154 |
| Table 14.3.1.2.3.2: Shift Table for Numeric Urinalysis Results (Safety Population) |
| Table 14.3.1.2.3.3: Summary of Character Urinalysis Results by Visit (Safety Population)155 |




Date: 24 MAY 2019

Table 14.0.1: Summary of Subject Completion/Discontinuation (Randomized Subjects)

| | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>Combined<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Completed Study | | | | | | | |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Reason for Discontinuation from Study | | | | | | | |
| Adverse Event | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) |
| Death | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost to Follow-Up | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Physician Decision | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pregnancy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Protocol Violation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Study Terminated by Sponsor | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Withdrawal by Subject | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Worsening Condition | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |




Date: 24 MAY 2019

Table 14.0.2: Summary of Subjects Excluded from Analyses (Randomized Subjects)

| Number of Subjects Included in the ITT Population | Vehicle QD (N=xx) xx (xx.x%) | Vehicle BID (N=xx) xx (xx.x%) | Vehicle<br>Combined<br>(N=xx)<br>xx (xx.x%) | BTX 1503<br>5% BID<br>(N=xx)<br>xx ( xx.x%) | BTX 1503<br>5% QD<br>(N=xx)<br>xx ( xx.x%) | BTX 1503<br>2.5% QD<br>(N=xx)<br>xx ( xx.x%) | BTX 1503<br>Combined<br>(N=xx)<br>xx (xx.x%) |
|---|---|---|---|---|---|---|---|
| Number of Subjects Included in the Safety Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded from the Safety Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Reason for Exclusion from the Safety Population | ( 0() | ( 0() | ( 0() | ( 0() | ( 0() | ( 0/) | ( 0/) |
| No Evidence of Subject Dosing | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | , | xx ( xx.x%) | 1 | xx ( xx.x%) |
| No Post Baseline Assessment | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Included in the PP Population<br>Number of Subjects Excluded from the PP Population<br>Reason for Exclusion from the PP Population | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) | | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |
| Violated the Inclusion/Exclusion Criteria | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Received an Interfering Medication | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Has not been Compliant with the Dosing Regimen | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missed IGA or Lesion Count assessment at Day 84 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missed Both Day 28 and Day 56 Visits | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Compliant with Dosing Regimen | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Day 84 Visit not within +/- 5 days Window | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other <sup>a</sup> | | | | | | | |

<sup>&</sup>lt;sup>a</sup> See Listing 16.2.3 for a complete list of all other reasons for exclusion from the PP population.

Note: ITT exclusion of not being randomized not presented due to requirement of needing to be randomized to be summarized in the table. Percentages are based on the number of randomized subjects.




Date: 24 MAY 2019

### Table 14.0.3: Summary of Reasons for Screen Failure (Non-Randomized Subjects)

| | Total<br>(N=xx) |
|-----------------------------------------------|-----------------|
| Reason for Screen Failure | |
| Adverse Event | xx ( xx.x%) |
| Inclusion and/or Exclusion Criteria | XX (XX.X%) |
| Withdrawal by Subject | xx ( xx.x%) |
| Withdrawal by Legally Authorized Representive | xx ( xx.x%) |
| Lost to Follow-Up | xx ( xx.x%) |
| Other | xx ( xx.x%) |

Note: Percentages are based on the number of non-randomized subjects.




Date: 24 MAY 2019

Table 14.1.1.1: Summary of Subject Demographics (ITT Population) 

| Age (years) | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>Combined<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx |
| Sex | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Male | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Female | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Ethnicity | | | | | | | |
| n<br>Hispanic or Latino<br>Not Hispanic or Latino | xx<br>xx ( xx.x%)<br>xx ( xx.x%) | xx<br>xx ( xx.x%)<br>xx ( xx.x%) | xx<br>xx ( xx.x%)<br>xx ( xx.x%) | | xx (xx.x%)<br>xx (xx.x%) | xx<br>xx ( xx.x%)<br>xx ( xx.x%) | xx<br>xx ( xx.x%)<br>xx ( xx.x%) |

Note: Percentages are based on the number of subjects in the ITT population with a non-missing response.




Date: 24 MAY 2019

Table 14.1.1.1: Summary of Subject Demographics (ITT Population) 

| | Vehicle QD (N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>Combined<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Race | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| American Indian or Alaska Native | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Asian | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Black or African American | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| White | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Multiple/Other | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Percentages are based on the number of subjects in the ITT population with a non-missing response.




Date: 24 MAY 2019

Repeat Table 14.1.1.1 for the following:

Table 14.1.1.2: Summary of Subject Demographics (PP Population)
Table 14.1.1.3: Summary of Subject Demographics (Safety Population)



otanix BTX.2018.001 Version: v1 Date: 24 MAY 2019

Table 14.1.2.1: Summary of Baseline Characteristics (ITT Population)


| Height (cm) | Vehicle QD (N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>Combined<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | xx, xx | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx |
| Weight (kg) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx |
| Alcohol History | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Drinker | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Non-drinker | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Smoking History | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Non-smoker | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Ex-smoker | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Smoker | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.1.2.1: Summary of Baseline Characteristics

(ITT Population)


| Lu Claurens de con Laciana Carret | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>Combined<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Inflammatory Lesion Count | | | | | | | |
| n<br>M | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Non-Inflammatory Lesion Count | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | xx, xx | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Total Lesion Count | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | XX, XX | xx, xx |




Date: 24 MAY 2019

Table 14.1.2.1: Summary of Baseline Characteristics (ITT Population) 

| | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>Combined<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Investigator Global Assessment | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.1.2.1 for the following:

Table 14.1.2.2: Summary of Baseline Characteristics (PP Population)
Table 14.1.2.3: Summary of Baseline Characteristics (Safety Population)




Date: 24 MAY 2019

Table 14.1.3.1: Summary of Concomitant Medications by ATC Level 2 Term and Preferred Name (ITT Population)

| ATC Level 2 Term Preferred Name <sup>a</sup> | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>Combined<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Subjects with at Least One Concomitant<br>Medication Reported | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ATC Level 2 Term 1 Preferred Name 1 Preferred Name 2 Preferred Name x | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

. . .

Note: Concomitant medications are those used on or after the date of first application of study medication. Percentages are based on the number of subjects in each treatment group in the ITT population. Subjects are only counted once per ATC Level 2 Term and once per Preferred Name.

<sup>&</sup>lt;sup>a</sup> WHO-DDE, Format B2, Version MAR 2017.




Date: 24 MAY 2019

Repeat Table 14.1.3.1 for the following:

Table 14.1.3.2: Summary of Concomitant Medications by ATC Level 2 Term and Preferred Name (PP Population) Table 14.1.3.3: Summary of Concomitant Medications by ATC Level 2 Term and Preferred Name (Safety Population)




Date: 24 MAY 2019

Table 14.1.4.1: Summary of Concomitant Antibiotic Therapies by ATC Level 2 Term and Preferred Name (ITT Population)

| ATC Level 2 Term Preferred Name <sup>a</sup> | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>Combined<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Subjects with at Least One Concomitant<br>Antibiotic Therapy Reported | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ATC Level 2 Term 1 Preferred Name 1 Preferred Name 2 Preferred Name x | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

. . .

Note: Concomitant antibiotic therapies are those used on or after the date of first application of study medication Percentages are based on the number of subjects in each treatment group in the ITT population. Subjects are only counted once per ATC Level 2 Term and once per Preferred Name.

<sup>&</sup>lt;sup>a</sup> WHO-DDE, Format B2, Version MAR 2017.




Date: 24 MAY 2019

Repeat Table 14.1.4.1 for the following:

Table 14.1.4.2: Summary of Concomitant Antibiotic Therapies by ATC Level 2 Term and Preferred Name (PP Population)

Table 14.1.4.3: Summary of Concomitant Antibiotic Therapies by ATC Level 2 Term and Preferred Name (Safety Population)




Date: 24 MAY 2019

Table 14.2.1.1: Primary Efficacy Endpoint: Summary of Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (ITT Population)

| Change from Baseline in<br>Inflammatory Lesion Counts | Vehicle QD<br>(N=xx) | Vehicle BID<br>(N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | Skewness<br>P-value |
|---|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| Min., Max. | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | |
| LSMeana | | | XX.X | XX.X | XX.X | XX.X | $0.xxxx^b$ |
| LSSDa | | | XX.XX | XX.XX | XX,XX | XX.XX | |
| Unranked P-value vs. Combined Vehicle <sup>a</sup> | | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Combined Vehicle <sup>c</sup> | | | | 0.xxxx | 0.xxxx | 0.xxxx | |

Note: Missing values imputed using LOCF.

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values from an analysis of covariance with factors of treatment group (vehicle treatment groups included as single combined treatment group) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>b</sup> Skewness test is based on methods presented by J.H. Zar (1984).

<sup>&</sup>lt;sup>c</sup> Contrast p-values from a ranked analysis of covariance with factors of treatment group (vehicle treatment groups included as single combined treatment group) and corresponding baseline lesion count as the covariate.




Date: 24 MAY 2019

Repeat Table 14.2.1.1 for the following:

Table 14.2.1.2: Primary Efficacy Endpoint: Summary of Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population) Programming note: replace last footnote with:

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Sensitivity Analysis of Primary Efficacy Endpoint: Summary of Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (ITT Population)

| Repeated Measures Analysis on Observed Data Change from Baseline in Inflammatory Lesion Counts | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| LSMean <sup>a</sup> | | | XX.X | XX.X | XX.X | XX.X |
| $LSSD^a$ | | | XX.XX | XX.XX | XX.XX | XX.XX |
| P-value vs. Combined Vehicle <sup>a</sup> | | | | 0.xxxx | 0.xxxx | 0.xxxx |

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values from a repeated measures analysis of covariance with factors of treatment group (vehicle treatment groups included as single combined treatment group), visit, treatment by visit interaction, and corresponding baseline lesion count as the covariate. Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| | | Baseli | ne Inflammatory l | Lesion Count < med | dian (xx) | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | , , | , , | | , , , | , , |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |
| | Baseline Inflammatory Lesion Count $\geq$ median (xx) | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| | | Baseline | Non-Inflammator | y Lesion Count < n | nedian (xx) | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | . , | , , , , | | , , | • | , , , |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | Baseline Non-Inflammatory Lesion Count $\geq$ median (xx) | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | N=xx | N=xx | (N=xx) | (N=xx) | N=xx | (N=xx) |
| Change from Baseline in | | | | | | |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| 3.61 | | | | | | |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| | | В | aseline Total Lesio | n Count < median | (xx) | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | | | | | , , , | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX,XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | Baseline Total Lesion Count $\geq$ median (xx) | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| TEXT 1 500 | 502 | DEN 1502 | | | | | |
|---|---|---|---|---|---|---|---|
| BTX 1503 | | BTX 1503 | BTX 1503 | Vehicle | W.1.1.1. DID | W.1.:.1. OD | |
| 2.5% QD | - | 5% QD | 5% BID | Combined | Vehicle BID | Vehicle QD | |
| (N=xx) | <u>X.)</u> | (N=xx) | (N=xx) | N=xx | (N=xx) | (N=xx) | |
| | | | | | | | Change from Baseline in<br>Inflammatory Lesion Counts |
| XX | XX | XX | XX | XX | XX | XX | n |
| XX.X | X.X | XX.X | XX.X | XX.X | XX.X | XX.X | Mean |
| XX.XX | .XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | SD |
| XX.X | X.X | XX.X | XX.X | XX.X | XX.X | XX.X | Median |
| XX, XX | XX | xx, xx | xx, xx | XX, XX | xx, xx | XX, XX | Min., Max. |
| BTX 1503 | 503 | BTX 1503 | A of 4 (Severe)<br>BTX 1503 | Vehicle | | | |
| 2.5% QD | D | 5% QD | 5% BID | Combined | Vehicle BID | Vehicle QD | |
| (N=xx) | - | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | |
| | | | | | | | Change from Baseline in |
| | | | | | | | Inflammatory Lesion Counts |
| XX | XX | XX | XX | XX | XX | XX | n |
| XX.X | X.X | XX.X | XX.X | XX.X | XX.X | XX.X | Mean |
| XX.XX | .XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | SD |
| XX.X | X.X | XX.X | XX.X | XX.X | XX.X | XX.X | Median |
| | vv | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | Min., Max. |
| | X.X<br>.XX<br>X.X | XX.X<br>XX.XX<br>XX.X | XX.X<br>XX.XX<br>XX.X | XX.X<br>XX.XX<br>XX.X | XX.XX<br>XX.X | XX.X<br>XX.XX<br>XX.X | Mean<br>SD<br>Median |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| | | Baseline A | .cne-OoL: Self-Per | ception Domain < | median (xxx) | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | N=xx | (N=xx) | N=xx | N=xx | (N=xx) | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | | | | | | , |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX,XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | Baseline Acne-QoL: Self-Perception Domain ≥ median (xxx) | | | | | |
| | W 11 1 OD | W. L. L. DID | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| | Baseline | Acne-OoL: Role-S | Social Domain < mo | edian (xxx) | |
|---|---|---|---|---|---|
| | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| (N=xx) | (N=xx) | (N=xx) | (N=xx) | | (N=xx) |
| | <u>, , </u> | | , | | , |
| XX | XX | XX | XX | XX | XX |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |
| Baseline Acne-QoL: Role-Social Domain ≥ median (xxx) Vehicle BTX 1503 BTX 1503 BTX 150 | | | | | |
| Vehicle OD | Vehicle BID | | | | 2.5% QD |
| • | | | | • | (N=xx) |
| XX | XX | XX | XX | XX | XX |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |
| | XX | Vehicle QD (N=xx) Vehicle BID (N=xx) xx xx xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx xx.x xx xx.x xx xx xx xx xx xx.x xx.x xx.x | Vehicle QD (N=xx) Vehicle BID (N=xx) Vehicle Combined (N=xx) XX XX XX XX XX.X XX.X XX.X XX.XX XX.X XX.XX XX.XX XX.XX XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX XX.X XX.X XX.X XX.X XX.X XX.X XX.X | $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Vehicle QD<br>(N=xx)Vehicle BID<br>(N=xx)Combined<br>(N=xx)5% BID<br>(N=xx)5% QD<br>(N=xx)xxxxxxxxxxxxxx.xxx.xxx.xxx.xxx.xxx.xxx.xxxx.xxxx.xxxx.xxxx.xxxx.xxxx.xxx.xxx.xxx.xxx.xxx.xxx.xxx.xxx.xxx.xxx.xxx.xxx.xxx.xxx.xxx.xxx.xxx.xVehicle QD<br>(N=xx)Vehicle BID<br>(N=xx)Combined<br>(N=xx)5% BID<br>(N=xx)5% QD<br>(N=xx)xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| | | Baseline A | cne-OoL: Role-En | notional Domain < | median (xxx) | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | N=xx | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | Baseline Acne-QoL: Role-Emotional Domain ≥ median (xxx) | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | , | | |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| | | Baselii | ne Acne-OoL: Acn | e Symptoms < med | ian (xxx) | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | N=xx | (N=xx) | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | , | | | | | , |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX,XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | Baseline Acne-QoL: Acne Symptoms ≥ median (xxx) | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| | | | DD C | | | |
|---|---|---|---|---|---|---|
| | | | | Improved | DEM 1500 | DEL 1500 |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | N=xx | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| | | | PRO | : Same | | |
| | | | PRO<br>Vehicle | <b>Same</b> BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | | | BTX 1503<br>5% QD | BTX 1503<br>2.5% QD |
| | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle | BTX 1503 | | |
| Change from Baseline in | | | Vehicle<br>Combined | BTX 1503<br>5% BID | 5% QD | 2.5% QD |
| Change from Baseline in<br>Inflammatory Lesion Counts | | | Vehicle<br>Combined | BTX 1503<br>5% BID | 5% QD | 2.5% QD |
| | | | Vehicle<br>Combined | BTX 1503<br>5% BID | 5% QD | 2.5% QD |
| <b>Inflammatory Lesion Counts</b> | (N=xx) | <u>(N=xx)</u> | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | 5% QD<br>(N=xx) | 2.5% QD<br>(N=xx) |
| Inflammatory Lesion Counts n | (N=xx) | (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | 5% QD<br>(N=xx) | 2.5% QD<br>(N=xx) |
| Inflammatory Lesion Counts<br>n<br>Mean | (N=xx) xx xx.x | (N=xx)<br>xx<br>xx.x | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | 5% QD<br>(N=xx)<br>xx<br>xx.x | 2.5% QD<br>(N=xx)<br>xx<br>xx.x |
| Inflammatory Lesion Counts n Mean SD | (N=xx) xx xx.x xx.x | XX XX.X XX.XX | Vehicle Combined (N=xx) xx xx.x xx.xx | BTX 1503 5% BID (N=xx) xx xx.x xx.xx | 5% QD<br>(N=xx)<br>xx<br>xx.x<br>xx.x | 2.5% QD<br>(N=xx)<br>xx<br>xx.x<br>xx.x |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| | PRO: Worsened | | | | | |
|---|---|---|---|---|---|---|
| | Vehicle BTX 1503 BTX 1503 | | | | | |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx | XX, XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| | | | | US | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | N=xx | (N=xx) | (N=xx) |
| Change from Baseline in | . , | | , | | | |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | | | 4 | AUS | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | N=xx | (N=xx) | N=xx | (N=xx) | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| 171111., 17111/1. | AA, AA | AA, AA | AA, AA | AA, AA | AA, AA | AA, AA |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| | Male | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | N=xx | N=xx | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX |
| | | | | emale | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| 11 | | | | | | |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX |
| Mean | XX.X | | | | | |
| Mean<br>SD | XX.X<br>XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| | | | Hienoni | c or Latino | | |
|---|---|---|---|---|---|---|
| | Vehicle QD | Vehicle BID | Vehicle<br>Combined | BTX 1503<br>5% BID | BTX 1503<br>5% QD | BTX 1503<br>2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | | <u> </u> | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx | XX, XX |
| | | | Non-Hispa | nic or Latino | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (NI) | (NI) | (NI) | (NI) |
| | (11 /1/1) | (11 AA) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | (I\ AA) | (IV AA) | <u>(N-XX)</u> | (N=XX) | <u>(N-xx)</u> | <u> (N-XX)</u> |
| | xx | XX | (N-xx) | (IN=XX) | (N-xx)xx | XX |
| Inflammatory Lesion Counts n Mean | , , | | · | | | |
| Inflammatory Lesion Counts n | xx | XX | xx | xx | xx | xx |
| Inflammatory Lesion Counts n Mean | XX<br>XX.X | xx<br>xx.x | XX<br>XX.X | xx<br>xx.x | xx<br>xx.x | xx<br>xx.x |
| Inflammatory Lesion Counts n Mean SD | XX<br>XX.X<br>XX.XX | XX<br>XX.X<br>XX.XX | XX<br>XX.X<br>XX.XX | XX<br>XX.X<br>XX.XX | XX<br>XX.X<br>XX.XX | XX<br>XX.X<br>XX.XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| | White | | | | | |
|---|---|---|---|---|---|---|
| | Vehicle QD | Vehicle BID | Vehicle<br>Combined | BTX 1503<br>5% BID | BTX 1503<br>5% QD | BTX 1503<br>2.5% QD |
| | (N=xx) | (N=xx) | N=xx | N=xx | (N=xx) | N=xx |
| Change from Baseline in Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX,XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx |
| | | | Non | -White | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | N=xx | (N=xx) | (N=xx) | (N=xx) | N=xx | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | , , | , , | | | , , | ` , |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| Vehicle QD (N=xx) xx xx.x | Vehicle BID (N=xx) xx | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|
| (N=xx) | <u>(N=xx)</u> | <u>(N=xx)</u> | | | • |
| xx | | , | <u>(N=xx)</u> | (N=xx) | <u>(N=xx)</u> |
| | xx | | | | |
| | XX | | | | |
| | XX | | | | |
| vv v | | XX | XX | XX | XX |
| ΛΛ.Λ | XX.X | XX.X | XX.X | XX.X | XX.X |
| XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| xx, xx | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |
| Age 18 to < 30 years | | | | | |
| | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| Vehicle OD | Vehicle BID | Combined | 5% BID | 5% OD | 2.5% QD |
| • | | | (N=xx) | | N=xx |
| | | | | | (= , ===, |
| XX | XX | XX | XX | XX | XX |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| XX, XX | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx |
| | Vehicle QD (N=xx) xx xx.x xx.x xx.x xx.xx xx.xx | xx.x xx.x xx, xx xx, xx Vehicle QD (N=xx) Vehicle BID (N=xx) xx xx xx xx xx.x xx.x xx.x xx.x | $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.3: Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population)


| | Age 30 to 40 years | | | | | |
|---|---|---|---|---|---|---|
| | Vehicle BTX 1503 BTX 1503 | | | | | |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.4: Responder Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population - Responders) 

| | | Baseli | ne Inflammatory I | Lesion Count < med | dian (xx) | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | N=xx | (N=xx) | (N=xx) |
| Change from Baseline in | | | . , | , | | |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| | Baseline Inflammatory Lesion Count $\geq$ median (xx) | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.




Table 14.2.1.4: Responder Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population - Responders)


| | | Baseline Non-Inflammatory Lesion Count < median (xx) | | | | |
|---|---|---|---|---|---|---|
| | | Buscinc | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | N=xx | (N=xx) | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |
| | Baseline Non-Inflammatory Lesion Count ≥ median (xx) | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| <b>Inflammatory Lesion Counts</b> | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.4: Responder Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population - Responders)


| | Baseline Total Lesion Count < median (xx) | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | , , | , , | , | | , | , , |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX,XX | XX.XX | XX,XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx |
| | | В | aseline Total Lesio | on Count ≥ median | (xx) | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in<br>Inflammatory Lesion Counts | , , | , , | , , | | , | , , |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.

 $SOURCE: USERNAME \verb|SPONSOR|| PROJECT \verb|JOBNAME|| (DATE, TIME)$ 




Table 14.2.1.4: Responder Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population - Responders)


| | | | Baseline IGA | of 3 (Moderate) | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | N=xx | N=xx | N=xx | (N=xx) | (N=xx) |
| Change from Baseline in | | | · | | | <u> </u> |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx |
| | | | Raseline IG | A of 4 (Severe) | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | **** | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | | |
| SD<br>Median | XX.XX<br>XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | | XX.X<br>XX, XX | XX.X<br>XX, XX | XX.X<br>XX, XX |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.1.4: Responder Subgroup Summary of the Primary Endpoint: Absolute Change from Baseline in Inflammatory Lesion Count at Day 84 (PP Population - Responders)


| | | | Percent Complian | ce < median (xx.x% | <b>6</b> ) | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | <del></del> | | | |
| Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| | | | | ce≥ median (xx.x% | <b>(6)</b> | |
| | | | Percent Complian<br>Vehicle | <b>ce ≥ median (xx.x%</b><br>BTX 1503 | 6)<br>BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | | • | * | BTX 1503<br>2.5% QD |
| | Vehicle QD<br>(N=xx) | | Vehicle | BTX 1503 | BTX 1503 | |
| Change from Baseline in | • | Vehicle BID | Vehicle<br>Combined | BTX 1503<br>5% BID | BTX 1503<br>5% QD | 2.5% QD |
| Change from Baseline in<br>Inflammatory Lesion Counts | • | Vehicle BID | Vehicle<br>Combined | BTX 1503<br>5% BID | BTX 1503<br>5% QD | 2.5% QD |
| | • | Vehicle BID | Vehicle<br>Combined | BTX 1503<br>5% BID | BTX 1503<br>5% QD | 2.5% QD |
| Inflammatory Lesion Counts | (N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | 2.5% QD<br>(N=xx) |
| Inflammatory Lesion Counts n | (N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | 2.5% QD<br>(N=xx) |
| Inflammatory Lesion Counts n Mean | XX XX.X | Vehicle BID (N=xx) xx xx.x | Vehicle Combined (N=xx) xx xx.x | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | 2.5% QD<br>(N=xx)<br>xx<br>xx.x |
| Inflammatory Lesion Counts n Mean SD | XX XX.X XX.XX | Vehicle BID (N=xx) xx xx.x xx.xx | Vehicle Combined (N=xx) xx xx.x xx.x | BTX 1503 5% BID (N=xx) xx xx.x xx.xx | BTX 1503 5% QD (N=xx) xx xx.x xx.xx | 2.5% QD<br>(N=xx)<br>xx<br>xx.x<br>xx.x |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.

 $SOURCE: USERNAME \verb|SPONSOR|| PROJECT \verb|JOBNAME|| (DATE, TIME)$ 




Date: 24 MAY 2019

Table 14.2.2.1.1: Secondary Efficacy Endpoint: Summary of Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (ITT Population)

| Change from Baseline in<br>Non-Inflammatory Lesion Counts | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | Skewness<br>P-value |
|---|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| Min., Max. | xx, xx | xx, xx | XX, XX | XX, XX | XX, XX | xx, xx | |
| LSMeana | | | XX.X | XX.X | XX.X | XX.X | $0.xxxx^b$ |
| LSSD <sup>a</sup> | | | XX.XX | XX.XX | XX.XX | XX.XX | |
| Unranked P-value vs. Combined Vehicle <sup>a</sup> | | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Combined Vehicle <sup>c</sup> | | | | 0.xxxx | 0.xxxx | 0.xxxx | |

Note: Missing values imputed using LOCF.

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values from an analysis of covariance with factors of treatment group (vehicle treatment groups included as single combined treatment group) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>b</sup> Skewness test is based on methods presented by J.H. Zar (1984).

<sup>&</sup>lt;sup>c</sup> Contrast p-values from a ranked analysis of covariance with factors of treatment group (vehicle treatment groups included as single combined treatment group) and corresponding baseline lesion count as the covariate.




Date: 24 MAY 2019

Repeat Table 14.2.2.1.1 for the following:

Table 14.2.2.1.2: Secondary Efficacy Endpoint: Summary of Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) *Programming note: replace last footnote with:* 

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.3: Sensitivity Analysis of Secondary Efficacy Endpoint: Summary of Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day

84

(ITT Population)

| Repeated Measures Analysis on Observed<br>Data<br>Change from Baseline in<br>Non-Inflammatory Lesion Counts | Vehicle QD (N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| LSMean <sup>a</sup><br>LSSD <sup>a</sup><br>P-value vs. Combined Vehicle <sup>a</sup> | | | XX.X<br>XX.XX | xx.x<br>xx.xx<br>0.xxxx | xx.x<br>xx.xx<br>0.xxxx | xx.x<br>xx.xx<br>0.xxxx |

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values from a repeated measures analysis of covariance with factors of treatment group (vehicle treatment groups included as single combined treatment group), visit, treatment by visit interaction, and corresponding baseline lesion count as the covariate. Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) 

| | Baseline Inflammatory Lesion Count < median (xx) | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | <del></del> _ | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| | | Baseli | ne Inflammatory I | Lesion Count ≥ med | lian (xx) | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | | | VV VV | XX.XX | VV VV | XX.XX |
| SD | XX.XX | XX.XX | XX.XX | λλ.λλ | XX.XX | ΛΛ.ΛΛ |
| Median | XX.XX<br>XX.X | XX.XX<br>XX.X | XX.XX<br>XX.X | XX.XX<br>XX.X | XX.XX<br>XX.X | XX.X |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) 

| | Baseline Non-Inflammatory Lesion Count < median (xx) | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | N=xx | (N=xx) | (N=xx) |
| Change from Baseline in<br>Non-Inflammatory Lesion Counts | | | | | | , |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx |
| | Baseline Non-Inflammatory Lesion Count ≥ median (xx) | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) 

| | Baseline Total Lesion Count < median (xx) | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | | В | aseline Total Lesio | n Count≥ median | (xx) | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | VV V | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | AA.A | | | | |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Note: No imputations were made for missing data.



Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) 

| | | | | of 3 (Moderate) | DELY 1502 | DEN. 1502 |
|---|---|---|---|---|---|---|
| | Vehicle QD | Vehicle BID | Vehicle<br>Combined | BTX 1503<br>5% BID | BTX 1503<br>5% QD | BTX 1503<br>2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | (1\ AA) | (IV AA) | (1\ AA) | <u> (11 AA)</u> | (1\ AA) | (1\ AA) |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx | XX, XX |
| | Baseline IGA of 4 (Severe) | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | N=xx | (N=xx) | (N=xx) |
| Change from Baseline in | , | | | | | <del> </del> |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| 1,1111., 1,111. | 11/1, /1/1 | 2222, 7272 | /1/1 /1/1 | 1111, 1111 | /1/1 <sub>1</sub> /1/1 | 71/1, 71/1 |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) 

| | | Baseline A | .cne-OoL: Self-Per | ception Domain < 1 | median (xxx) | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | | Baseline A | .cne-QoL: Self-Per | ception Domain≥ | median (xxx) | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | N=xx | <u>(N=xx)</u> | N=xx | (N=xx) | N=xx | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | | | , | , | , | , |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population)


| | | Baseline | Acne-OoL: Role-S | Social Domain < mo | edian (xxx) | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in<br>Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | xx, xx | xx, xx | XX, XX | XX, XX | xx, xx |
| | Baseline Acne-QoL: Role-Social Domain ≥ median (xxx) | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | , | , | , | , | , | , |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population)


Baseline Acne-QoL: Role-Emotional Domain < median (xxx) Vehicle BTX 1503 BTX 1503 BTX 1503 Combined 5% QD 2.5% QD Vehicle OD Vehicle BID 5% BID (N=xx)(N=xx)(N=xx)(N=xx)(N=xx)(N=xx)**Change from Baseline in Non-Inflammatory Lesion Counts** XXXXXXXXXXXXMean XX.X XX.X XX.X XX.X XX.XXX.X SD XX.XX XX.XX XX.XX XX.XXXX.XX XX.XX Median XX.X XX.X XX.X XX.X XX.XXX.X Min., Max. XX, XX XX, XX XX, XX XX, XX XX, XX XX, XX Baseline Acne-QoL: Role-Emotional Domain ≥ median (xxx) Vehicle BTX 1503 BTX 1503 BTX 1503 Vehicle QD Vehicle BID Combined 5% BID 5% QD 2.5% QD (N=xx)(N=xx)(N=xx)(N=xx)(N=xx)(N=xx)**Change from Baseline in Non-Inflammatory Lesion Counts** n XXXXXXXXXXXXMean XX.X XX.XXX.XXX.X XX.X XX.X SD XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX Median XX.XXX.XXX.X XX.X XX.XXX.X Min., Max. XX, XX XX, XX XX, XX XX, XX XX, XX XX, XX

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) 

| | | Baselii | ne Acne-OoL: Acn | e Symptoms < med | ian (xxx) | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in<br>Non-Inflammatory Lesion Counts | | , , | , | | , , | , , , |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx |
| | Baseline Acne-QoL: Acne Symptoms ≥ median (xxx) | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) 

| | PRO: Improved | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | N=xx | (N=xx) | (N=xx) |
| Change from Baseline in | | , , | , , | , , , | , , | , , |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx |
| | | | DD.C | ): Same | | |
| | | | Vehicle | BTX 1503 | DTV 1502 | DTV 1502 |
| | | | venicie | D1A 1303 | BTX 1503 | BTX 1503 |
| | Walsiala OD | Walsiala DID | | | 50/ OD | 2.50/ OD |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | | | 5% QD<br>(N=xx) | 2.5% QD<br>(N=xx) |
| Change from Baseline in<br>Non-Inflammatory Lesion Counts | | | Combined | 5% BID | • | - |
| | | | Combined | 5% BID | • | - |
| Non-Inflammatory Lesion Counts | (N=xx) | <u>(N=xx)</u> | Combined<br>(N=xx) | 5% BID<br>(N=xx) | (N=xx) | (N=xx) |
| Non-Inflammatory Lesion Counts<br>n | (N=xx) | (N=xx) | Combined<br>(N=xx) | 5% BID<br>(N=xx) | (N=xx) | (N=xx) |
| Non-Inflammatory Lesion Counts<br>n<br>Mean | (N=xx) xx xx.x | (N=xx) xx xx.x | Combined (N=xx) xx xx.x | 5% BID<br>(N=xx)<br>xx<br>xx.x | (N=xx) xx xx.x | (N=xx) xx xx.x |
| Non-Inflammatory Lesion Counts n Mean SD | (N=xx)<br>xx<br>xx.x<br>xx.x | XX XX.X XX.XX | Combined (N=xx) xx xx.x xx.x | 5% BID<br>(N=xx)<br>xx<br>xx.x<br>xx.x | (N=xx)<br>xx<br>xx.x<br>xx.x | (N=xx) xx xx.x xx.xx |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) 

| | PRO: Worsened | | | | | |
|---|---|---|---|---|---|---|
| | Vehicle BTX 1503 BTX 1503 | | | | | |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | N=xx | (N=xx) | (N=xx) | N=xx | N=xx | N=xx |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx | XX, XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) 

| | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | US BTX 1503 5% BID (N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| Change from Baseline in Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle Combined (N=xx) | AUS BTX 1503 5% BID (N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
| Change from Baseline in<br>Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx | XX, XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) 

| | | | N<br>Vehicle | Male<br>BTX 1503 | BTX 1503 | BTX 1503 |
|---|---|---|---|---|---|---|
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | N=xx | (N=xx) | N=xx | N=xx | N=xx | (N=xx) |
| Change from Baseline in<br>Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX,XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |
| | | | Fe | emale | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Mean<br>SD | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) 

| | Hispanic or Latino | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | | | | nic or Latino | | |
| | | | ** 1 1 1 | DTX 1503 | DTX 1500 | DTV 1502 |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Vehicle<br>Combined | 5% BID | 5% QD | 2.5% QD |
| | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | | | | |
| Change from Baseline in | | | Combined | 5% BID | 5% QD | 2.5% QD |
| Change from Baseline in<br>Non-Inflammatory Lesion Counts | | | Combined | 5% BID | 5% QD | 2.5% QD |
| | | | Combined | 5% BID | 5% QD | 2.5% QD |
| Non-Inflammatory Lesion Counts<br>n<br>Mean | (N=xx) | <u>(N=xx)</u> | Combined<br>(N=xx) | 5% BID<br>(N=xx) | 5% QD<br>(N=xx) | 2.5% QD<br>(N=xx) |
| Non-Inflammatory Lesion Counts<br>n | (N=xx) | (N=xx) | Combined<br>(N=xx) | 5% BID<br>(N=xx) | 5% QD<br>(N=xx) | 2.5% QD<br>(N=xx) |
| Non-Inflammatory Lesion Counts<br>n<br>Mean | (N=xx) xx xx.x | (N=xx) xx xx.x | Combined (N=xx) xx xx.x | 5% BID (N=xx) xx xx.x | 5% QD<br>(N=xx)<br>xx<br>xx.x | 2.5% QD<br>(N=xx)<br>xx<br>xx.x |
| Non-Inflammatory Lesion Counts n Mean SD | (N=xx) xx xx.x xx.x | XX XX.X XX.XX | Combined (N=xx) xx xx.x xx.x | 5% BID<br>(N=xx)<br>xx<br>xx.x<br>xx.x | 5% QD<br>(N=xx)<br>xx<br>xx.x<br>xx.x | 2.5% QD<br>(N=xx)<br>xx<br>xx.x<br>xx.x |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) 

| | White | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | N=xx | N=xx | (N=xx) | (N=xx) | N=xx | N=xx |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx |
| | | | Non | -White | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | | V.1.1.1. DID | | | | |
| | Vahiala OD | | L'amhinad | | | |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD<br>(N=vv) | 2.5% QD |
| Changa from Rasalina in | Vehicle QD<br>(N=xx) | (N=xx) | (N=xx) | (N=xx) | 5% QD<br>(N=xx) | 2.5% QD<br>(N=xx) |
| Change from Baseline in<br>Non-Inflammatory Lesion Counts | | | | | • | |
| | | | | | • | |
| Non-Inflammatory Lesion Counts<br>n<br>Mean | (N=xx) | (N=xx) | (N=xx) | <u>(N=xx)</u> | (N=xx) | (N=xx) |
| Non-Inflammatory Lesion Counts<br>n | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Non-Inflammatory Lesion Counts<br>n<br>Mean | (N=xx) xx xx.x | XX XX.X | XX XX.X | (N=xx) xx xx.x | (N=xx) xx xx.x | (N=xx) xx xx.x |
| Non-Inflammatory Lesion Counts n Mean SD | | XX XX.X XX.XX | XX XX.X XX.XX | XX XX.X XX.XX | (N=xx)<br>xx<br>xx.x<br>xx.x | (N=xx) xx xx.x xx.x |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population) 

| | Age 12 to < 18 years | | | | | |
|---|---|---|---|---|---|---|
| | Vehicle QD<br>(N=xx) | Vehicle BID<br>(N=xx) | Vehicle Combined (N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
| Change from Baseline in | (IV-XX) | $(1\sqrt{-\lambda\lambda})$ | (N-XX) | <u>(IV=XX)</u> | (IV-XX) | <u>(11–XX)</u> |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | xx, xx | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| | Age 18 to < 30 years | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | , , , , , , | , | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.4: Subgroup Summary of Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population)


| | Age 30 to 40 years | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | , , , | , , , | , , , |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.5: Responder Subgroup Summary of the Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84

(PP Population - Responders) 

| | | Baseli | ne Inflammatory I | Lesion Count < med | lian (xx) | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | Baseline Inflammatory Lesion Count $\geq$ median (xx) | | | | | |
| | | Duscii | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.




Date: 24 MAT 2019

Day 84 (PP Population - Responders) 

Table 14.2.2.1.5: Responder Subgroup Summary of the Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at

| | Baseline Non-Inflammatory Lesion Count < median (xx) | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX,XX | XX.XX | XX,XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx |
| | Baseline Non-Inflammatory Lesion Count $\geq$ median (xx) | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | N=xx | (N=xx) | (N=xx) |
| Change from Baseline in | | | | , | | , |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.1.5: Responder Subgroup Summary of the Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (PP Population - Responders) 

| | | В | aseline Total Lesio | on Count < median | (xx) | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| | Baseline Total Lesion Count $\geq$ median (xx) | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | N=xx | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | , |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.




Table 14.2.2.1.5: Responder Subgroup Summary of the Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at

Day 84

(PP Population - Responders)


| | | | | of 3 (Moderate) | DTV 1702 | DTV 1502 |
|---|---|---|---|---|---|---|
| | Vehicle QD | Vehicle BID | Vehicle<br>Combined | BTX 1503<br>5% BID | BTX 1503<br>5% QD | BTX 1503<br>2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | (1\ AA) | $\underline{\qquad}$ | $\frac{11 \Lambda \Lambda}{1}$ | (IV AA) | (11 AA) | (11 AA) |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx |
| | | | <b>D</b> 11 10 | | | |
| | | | | A of 4 (Severe) | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| | xx | XX | XX | XX | XX | xx |
| Non-Inflammatory Lesion Counts | XX<br>XX.X | XX<br>XX.X | XX<br>XX.X | XX<br>XX.X | XX<br>XX.X | XX<br>XX.X |
| Non-Inflammatory Lesion Counts<br>n | | | | | | |
| Non-Inflammatory Lesion Counts<br>n<br>Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Non-Inflammatory Lesion Counts<br>n<br>Mean<br>SD | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.




Table 14.2.2.1.5: Responder Subgroup Summary of the Secondary Efficacy Endpoint: Absolute Change from Baseline in Non-Inflammatory Lesion Count at
Day 84

(PP Population - Responders)


| | | | Percent Complian | ce < median (xx.x% | <b>(6)</b> | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | | | | | | |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| | Percent Compliance ≥ median (xx.x%) | | | | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Change from Baseline in | (1, 1212) | (1, 1111) | (1, 121) | (1, 121) | (1, 111) | (1, 1111) |
| Non-Inflammatory Lesion Counts | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.2.1: Secondary Efficacy Endpoint: Summary of Percent Change from Baseline in Inflammatory and Non-Inflammatory Lesion Count at Day 84 (ITT Population) 

| Percent Change from Baseline in<br>Inflammatory Lesion Counts | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | Skewness<br>P-value |
|---|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| Min., Max. | XX, XX | xx, xx | XX, XX | XX, XX | xx, xx | xx, xx | |
| LSMean <sup>a</sup> | | | XX.X | XX.X | XX.X | XX.X | $0.xxxx^b$ |
| $LSSD^a$ | | | XX.XX | XX.XX | XX.XX | XX.XX | |
| Unranked P-value vs. Combined Vehicle <sup>a</sup> | | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Combined Vehicle <sup>c</sup> | | | | 0.xxxx | 0.xxxx | 0.xxxx | |

Note: Missing values imputed using LOCF.

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values from an analysis of covariance with factors of treatment group (vehicle treatment groups included as single combined treatment group) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>b</sup> Skewness test is based on methods presented by J.H. Zar (1984).

<sup>&</sup>lt;sup>c</sup> Contrast p-values from a ranked analysis of covariance with factors of treatment group (vehicle treatment groups included as single combined treatment group) and corresponding baseline lesion count as the covariate.




Table 14.2.2.2.1: Secondary Efficacy Endpoint: Summary of Percent Change from Baseline in Inflammatory and Non-Inflammatory Lesion Count at Day 84 (ITT Population)


| Percent Change from Baseline in<br>Non-Inflammatory Lesion Counts | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | Skewness<br>P-value |
|---|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| Min., Max. | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | XX, XX | |
| LSMean <sup>a</sup> LSSD <sup>a</sup> Unranked P-value vs. Combined Vehicle <sup>a</sup> Ranked P-value vs. Combined Vehicle <sup>c</sup> | | | XX.X<br>XX.XX | xx.x<br>xx.xx<br>0.xxxx<br>0.xxxx | xx.x<br>xx.xx<br>0.xxxx<br>0.xxxx | xx.x<br>xx.xx<br>0.xxxx<br>0.xxxx | 0.xxxx <sup>b</sup> |

Note: Missing values imputed using LOCF.

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values from an analysis of covariance with factors of treatment group (vehicle treatment groups included as single combined treatment group) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>b</sup> Skewness test is based on methods presented by J.H. Zar (1984).

<sup>&</sup>lt;sup>c</sup> Contrast p-values from a ranked analysis of covariance with factors of treatment group (vehicle treatment groups included as single combined treatment group) and corresponding baseline lesion count as the covariate.




Date: 24 MAY 2019

Repeat Table 14.2.2.2.1 for the following:

Table 14.2.2.2.2: Secondary Efficacy Endpoint: Summary of Percent Change from Baseline in Inflammatory and Non-Inflammatory Lesion Count at Day 84 (PP Population)

Programming note: replace last footnote with:

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.1: Secondary Efficacy Endpoint: Summary of Dichotomized IGA at Day 84 (ITT Population)

| >= 2 Grade Reduction from Baseline in IGA<br>Success<br>Failure<br>P-value vs. Combined Vehicle <sup>a</sup> | Vehicle QD<br>(N=xx)<br>xx.x%<br>xx.x% | Vehicle BID (N=xx) xx.x% xx.x% | Vehicle<br>Combined<br>(N=xx)<br>xx.x%<br>xx.x% | BTX 1503<br>5% BID<br>(N=xx)<br>xx.x%<br>xx.x%<br>0.xxxx | BTX 1503<br>5% QD<br>(N=xx)<br>xx.x%<br>xx.x%<br>0.xxxx | BTX 1503<br>2.5% QD<br>(N=xx)<br>xx.x%<br>xx.x%<br>0.xxxx | Treatment P-value 0.xxxxa |
|---|---|---|---|---|---|---|---|
| IGA Grade of 0 or 1 Success Failure P-value vs. Combined Vehicle <sup>a</sup> | xx.x%<br>xx.x% | xx.x%<br>xx.x% | xx.x%<br>xx.x% | xx.x%<br>xx.x%<br>0.xxxx | xx.x%<br>xx.x%<br>0.xxxx | xx.x%<br>xx.x%<br>0.xxxx | 0.xxxx <sup>a</sup> |
| >= 2 Grade Reduction from Baseline and<br>IGA Grade of 0 or 1<br>Success<br>Failure<br>P-value vs. Combined Vehicle <sup>a</sup> | xx.x%<br>xx.x% | xx.x%<br>xx.x% | xx.x%<br>xx.x% | xx.x%<br>xx.x%<br>0.xxxx | xx.x%<br>xx.x%<br>0.xxxx | xx.x%<br>xx.x%<br>0.xxxx | 0.xxxx <sup>a</sup> |

<sup>&</sup>lt;sup>a</sup> P-value from a logistic regression with factor of treatment group (vehicle treatment groups included as single combined treatment group). Note: Missing values imputed using LOCF.




Date: 24 MAY 2019

Repeat Table 14.2.2.3.1 for the following:

Table 14.2.2.3.2: Secondary Efficacy Endpoint: Summary of Dichotomized IGA at Day 84 (PP Population)

Programming note: replace last footnote with:

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population) 

| | Baseline Inflammatory Lesion Count < median (xx) | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | | | | | | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | XX.X% | $XX.X^{0}/_{0}$ | XX.X% | xx.x% | XX.X% |
| Failure | XX.X% | xx.x% | XX.X% | XX.X% | xx.x% | XX.X% |
| | | Baseli | ne Inflammatory I | Lesion Count≥ med | lian (xx) | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | | | | | | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | XX.X% | $XX.X^{0}/_{0}$ | XX.X% | xx.x% | XX.X% |
| Failure | XX.X% | xx.x% | $XX.X^{0}/_{0}$ | XX.X% | xx.x% | xx.x% |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population) 

| Baseline Non-Inflammatory Lesion Count < median (xx) | | | | | |
|---|---|---|---|---|---|
| | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| N=xx | N=xx | (N=xx) | (N=xx) | N=xx | N=xx |
| xx.x% | XX.X% | xx.x% | XX.X% | xx.x% | XX.X% |
| XX.X% | XX.X% | xx.x% | XX.X% | XX.X% | XX.X% |
| | Baseline | Non-Inflammator | y Lesion Count≥ m | nedian (xx) | |
| | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| XX.X% | xx.x% | xx.x% | xx.x% | XX.X% | xx.x% |
| XX.X% | XX.X% | xx.x% | xx.x% | xx.x% | XX.X% |
| | XX.X% XX.X% Vehicle QD (N=xx) XX.X% | Vehicle QD (N=xx) XX.x% XX.x% XX.x% Baseline Vehicle QD (N=xx) Vehicle BID (N=xx) XX.x% XX.x% XX.x% XX.x% | Vehicle QD<br>(N=xx)Vehicle BID<br>(N=xx)Combined<br>(N=xx) $xx.x\%$<br>$xx.x\%$ $xx.x\%$<br>$xx.x\%$ $xx.x\%$<br>$xx.x\%$ Baseline Non-Inflammator<br>VehicleVehicle QD<br>(N=xx)Vehicle BID<br>(N=xx)Combined<br>(N=xx) $xx.x\%$ $xx.x\%$ | Vehicle QD<br>(N=xx)Vehicle BID<br>(N=xx)Vehicle Combined<br>(N=xx)BTX 1503<br>5% BID<br>(N=xx)xx.x%<br>xx.x%xx.x%<br>xx.x%xx.x%<br>xx.x%xx.x%<br>xx.x%Baseline Non-Inflammatory Lesion Count ≥ m<br>Vehicle<br>BTX 1503Vehicle QD<br>(N=xx)Vehicle BID<br>(N=xx)Combined<br>(N=xx)5% BID<br>(N=xx)xx.x%xx.x%xx.x% | Vehicle QD (N=xx) Vehicle BID (N=xx) Vehicle BID (N=xx) BTX 1503 (N=xx) BTX 1503 (N=xx) xx.x% xx.x% xx.x% xx.x% xx.x% xx.x% xx.x% xx.x% xx.x% xx.x% xx.x% Baseline Non-Inflammatory Lesion Count ≥ median (xx) Vehicle QD (N=xx) Vehicle BID (N=xx) Nempton Single |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population)


| | Baseline Total Lesion Count < median (xx) | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | | | | | | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | XX.X% | xx.x% | XX.X% | xx.x% | xx.x% |
| Failure | XX.X% | xx.x% | xx.x% | XX.X% | xx.x% | xx.x% |
| | | В | aseline Total Lesio | n Count ≥ median | (xx) | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 60/ DID | 50/ OD | 2.50/ OD |
| | V CHICLE QD | V CHICLE DID | Combined | 5% BID | 3% QD | 2.5% QD |
| | (N=xx) | | (N=xx) | 5% BID<br>(N=xx) | 5% QD<br>(N=xx) | 2.5% QD<br>(N=xx) |
| >= 2 Grade Reduction from Baseline and | - | (N=xx) | | | - | |
| >= 2 Grade Reduction from Baseline and IGA Grade of 0 or 1 | - | | | | - | |
| IGA Grade of 0 or 1 | - | | | | - | |
| IGA Grade of 0 or 1<br>Success | (N=xx)<br>xx.x% | (N=xx)<br>xx.x% | (N=xx)<br>xx.x% | (N=xx)<br>xx.x% | (N=xx)<br>xx.x% | (N=xx)<br>xx.x% |
| IGA Grade of 0 or 1 | (N=xx) | (N=xx) | <u>(N=xx)</u> | (N=xx) | (N=xx) | (N=xx) |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population) 

| >= 2 Grade Reduction from Baseline and | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Baseline IGA Vehicle Combined (N=xx) | of 3 (Moderate) BTX 1503 5% BID (N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | XX.X% |
| Failure | xx.x% | $XX.X^{0}/_{0}$ | XX.X% | $XX.X^{0}/_{0}$ | XX.X% | $XX.X^{0}/_{0}$ |
| | | | <b>Baseline IG</b> Vehicle | A of 4 (Severe)<br>BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and IGA Grade of 0 or 1 | (14-34) | <u> (IV-AA)</u> | (IV=XX) | (IV-AA) | (IV-XX) | <u> (IV-AA)</u> |
| Success | XX.X% | XX.X% | XX.X% | xx.x% | XX.X% | XX.X% |
| Failure | xx.x% | XX.X% | XX.X% | xx.x% | xx.x% | XX.X% |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population) 

| | Baseline Acne-QoL: Self-Perception Domain < median (xxx) | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | | | | | | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | $XX.X^{0}/_{0}$ | xx.x% | XX.X% | xx.x% | $XX.X^{0}/_{0}$ |
| Failure | xx.x% | XX.X% | XX.X% | XX.X% | xx.x% | XX.X% |
| | | Baseline A | cne-QoL: Self-Per | ception Domain≥ r | nedian (xxx) | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | | | | | | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | XX.X% | XX.X% | XX.X% | xx.x% | XX.X% |
| Failure | XX.X% | $XX.X^{0}/_{0}$ | $XX.X^{0}/_{0}$ | $XX.X^{0}/_{0}$ | XX.X% | $XX.X^{0}/_{0}$ |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population) 

| | Baseline Acne-QoL: Role-Social Domain < median (xxx) | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | | | | · | | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | XX.X% | xx.x% | XX.X% | XX.X% | XX.X% |
| Failure | xx.x% | XX.X% | xx.x% | XX.X% | XX.X% | XX.X% |
| | | Baseline | Acne-QoL: Role-S | Social Domain≥ me | edian (xxx) | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | , | | | | | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | XX.X% | XX.X% | xx.x% | xx.x% | XX.X% |
| Failure | xx.x% | XX.X% | XX.X% | XX.X% | xx.x% | xx.x% |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population) 

| Baseline Acne-QoL: Role-Emotional Domain < median (xxx) | | | | | |
|---|---|---|---|---|---|
| | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| | | | · | | |
| xx.x% | $xx.x^{0}/_{0}$ | xx.x% | xx.x% | XX.X% | $xx.x^{0}/_{0}$ |
| xx.x% | $XX.X^{0}/_{0}$ | xx.x% | $xx.x^{0}/_{0}$ | xx.x% | $XX.X^{0}/_{0}$ |
| | Baseline A | cne-QoL: Role-En | notional Domain≥ | median (xxx) | |
| | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| (N=xx) | N=xx | N=xx | (N=xx) | (N=xx) | (N=xx) |
| | | | | , | |
| xx.x% | xx.x% | xx.x% | xx.x% | $xx.x^{0}/_{0}$ | xx.x% |
| xx.x% | $XX.X^{0}/_{0}$ | xx.x% | xx.x% | XX.X% | $XX.X^{0}/_{0}$ |
| | XX.x% XX.x% Vehicle QD (N=xx) XX.x% | Vehicle QD (N=xx) Vehicle BID (N=xx) xx.x% xx.x% xx.x% xx.x% Baseline A Vehicle QD (N=xx) Vehicle BID (N=xx) xx.x% xx.x% | Vehicle QD<br>(N=xx)Vehicle BID<br>(N=xx)Combined<br>(N=xx) $xx.x\%$<br>$xx.x\%$ $xx.x\%$<br>$xx.x\%$ $xx.x\%$<br>$xx.x\%$ Baseline Acne-QoL: Role-En<br>Vehicle QD<br>(N=xx)Vehicle BID<br>(N=xx)Combined<br>(N=xx) $xx.x\%$ $xx.x\%$ $xx.x\%$ | $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Vehicle QD (N=xx) Vehicle BID (N=xx) Vehicle BID (N=xx) Vehicle BID (N=xx) BTX 1503 SW QD (N=xx) xx.x% xx.x% xx.x% xx.x% xx.x% xx.x% xx.x% xx.x% xx.x% xx.x% xx.x% xx.x% xx.x% Baseline Acne-QoL: Role-Emotional Domain ≥ median (xxx) Vehicle QD (N=xx) Vehicle BID (N=xx) N=xx N=xx Vehicle QD (N=xx) (N=xx) (N=xx) (N=xx) |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population) 

| Baseline Acne-QoL: Acne Symptoms < median (xxx) | | | | | |
|---|---|---|---|---|---|
| | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| N=xx | N=xx | (N=xx) | N=xx | (N=xx) | (N=xx) |
| xx.x% | XX.X% | xx.x% | xx.x% | XX.X% | XX.X% |
| XX.X% | xx.x% | xx.x% | xx.x% | XX.X% | XX.X% |
| | Baselir | ne Acne-QoL: Acn | e Symptoms ≥ medi | ian (xxx) | |
| | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | N=xx |
| xx.x% | XX.X% | xx.x% | xx.x% | XX.X% | XX.X% |
| XX.X% | xx.x% | xx.x% | xx.x% | XX.X% | XX.X% |
| | XX.X% XX.X% Vehicle QD (N=xx) XX.X% | Vehicle QD (N=xx) Vehicle BID (N=xx) xx.x% xx.x% xx.x% xx.x% Baselin Vehicle QD (N=xx) Vehicle BID (N=xx) xx.x% xx.x% | Vehicle QD<br>(N=xx)Vehicle BID<br>(N=xx)Combined<br>(N=xx) $xx.x\%$<br>$xx.x\%$ $xx.x\%$<br>$xx.x\%$ $xx.x\%$<br>$xx.x\%$ Baseline Acne-QoL: Acne-Vehicle<br>Vehicle QD<br>(N=xx)Vehicle BID<br>(N=xx)Combined<br>(N=xx) $xx.x\%$ $xx.x\%$ | Vehicle QD<br>(N=xx)Vehicle BID<br>(N=xx)Vehicle Combined<br>(N=xx)BTX 1503<br>5% BID<br>(N=xx)xx.x%<br>xx.x%xx.x%<br>xx.x%xx.x%<br>xx.x%xx.x%<br>xx.x%Baseline Acne-QoL: Acne Symptoms ≥ medical Vehicle<br>Vehicle QD<br>(N=xx)Vehicle BID<br>(N=xx)Combined<br>(N=xx)5% BID<br>(N=xx)xx.x%xx.x%xx.x% | Vehicle QD (N=xx) Vehicle BID (N=xx) Vehicle BID (N=xx) BTX 1503 (N=x) BTX 1503 (N=xx) XX.x% XX.x% |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population)


| | | | PDO. | Improved | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | N=xx | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | | | | | | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | XX.X% | XX.X% | xx.x% | XX.X% | XX.X% | XX.X% |
| Failure | xx.x% | XX.X% | XX.X% | XX.X% | XX.X% | xx.x% |
| | | | PRO | ): Same | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | N=xx | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | | | | | | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | XX.X% | xx.x% | XX.X% | XX.X% | XX.X% |
| Failure | XX.X% | XX.X% | xx.x% | XX.X% | XX.X% | XX.X% |
| | | | PRO: ' | Worsened | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | N=xx | N=xx | (N=xx) | (N=xx) | N=xx |
| >= 2 Grade Reduction from Baseline and | | | | | | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | XX.X% | XX.X% | XX.X% | $XX.X^{0}/_{0}$ | XX.X% | XX.X% |
| Failure | xx.x% | XX.X% | XX.X% | XX.X% | xx.x% | XX.X% |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population)


| >= 2 Grade Reduction from Baseline and | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | xx.x% | XX.X% | XX.X% | XX.X% | xx.x% |
| Failure | XX.X% | XX.X% | xx.x% | $XX.X^{0}/_{0}$ | XX.X% | XX.X% |
| | | | A | AUS | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and IGA Grade of 0 or 1 | | · | · | <del> </del> | · | · · · · · · |
| Success | xx.x% | $XX.X^{0}/_{0}$ | XX.X% | XX.X% | xx.x% | XX.X% |
| Failure | XX.X% | xx.x% | xx.x% | xx.x% | xx.x% | XX.X% |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population) 

| >= 2 Grade Reduction from Baseline and | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | Male BTX 1503 5% BID (N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| IGA Grade of 0 or 1 | | | | | | |
| Success | XX.X% | xx.x% | xx.x% | $XX.X^{0}/_{0}$ | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | $XX.X^{0}/_{0}$ | XX.X% | xx.x% | XX.X% |
| | | | Fe<br>Vehicle | emale<br>BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and IGA Grade of 0 or 1 | | | | | _(1\ 1112) | |
| Success | XX.X% | XX.X% | XX.X% | XX.X% | XX.X% | $XX.X^{0}/_{0}$ |
| Failure | xx.x% | $XX.X^{0}/_{0}$ | XX.X% | XX.X% | xx.x% | XX.X% |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population) 

| >= 2 Grade Reduction from Baseline and | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Hispanic<br>Vehicle<br>Combined<br>(N=xx) | c or Latino BTX 1503 5% BID (N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| IGA Grade of 0 or 1 | | | | | | |
| Success | XX.X% | XX.X% | xx.x% | xx.x% | XX.X% | $XX.X^{0}/_{0}$ |
| Failure | xx.x% | XX.X% | XX.X% | XX.X% | xx.x% | XX.X% |
| | Non-Hispanic or Latino Vehicle BTX 1503 BTX 1503 BTX 1503 | | | | | |
| | | 77 1 1 1 DTD | ~ 1. 1 | 50 / DID | 50/ OD | |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | Vehicle QD<br>(N=xx) | | | 5% BID<br>(N=xx) | 5% QD<br>(N=xx) | 2.5% QD<br>(N=xx) |
| >= 2 Grade Reduction from Baseline and IGA Grade of 0 or 1 | (N=xx) | <u>(N=xx)</u> | (N=xx) | (N=xx) | (N=xx) | <u>(N=xx)</u> |
| IGA Grade of 0 or 1<br>Success | (N=xx)<br>xx.x% | (N=xx)<br>xx.x% | (N=xx)<br>xx.x% | (N=xx)<br>xx.x% | (N=xx)<br>xx.x% | (N=xx)<br>xx.x% |
| IGA Grade of 0 or 1 | (N=xx) | <u>(N=xx)</u> | (N=xx) | (N=xx) | (N=xx) | <u>(N=xx)</u> |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population) 

| >= 2 Grade Reduction from Baseline and | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | /hite<br>BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | XX.X <sup>0</sup> / <sub>0</sub> | XX.X% | XX.X <sup>0</sup> / <sub>0</sub> | XX.X% | $XX.X^{0}/_{0}$ |
| Failure | xx.x% | $XX.X^{0}/_{0}$ | XX.X% | XX.X% | XX.X% | XX.X% |
| | | | Non | -White | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | XX.X% | XX.X% | XX.X% | XX.X% | xx.x% |
| Failure | xx.x% | XX.X% | XX.X% | XX.X% | XX.X% | xx.x% |

Note: No imputations were made for missing data.



Date: 24 MAY 2019

Table 14.2.2.3.3: Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population)


| | | | . 12. | . 10 | | |
|---|---|---|---|---|---|---|
| | | | Age 12 to<br>Vehicle | o < <b>18 years</b><br>BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | (1, 1111) | (1, 121) | (1, 1111) | (1, 121) | (1, 1111) | (1, 1111) |
| IGA Grade of 0 or 1 | | | | | | |
| Success | XX.X% | $XX.X^{0}/_{0}$ | xx.x% | $xx.x^{0}/_{0}$ | xx.x% | XX.X% |
| Failure | xx.x% | XX.X% | xx.x% | XX.X% | XX.X% | xx.x% |
| | | | A 10 4s | × 20 | | |
| | | | Vehicle | 0 < <b>30 years</b><br>BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | (11-77) | (11-XX) | (11-XX) | (1V-XX) | (11-77) | (11-XX) |
| IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | xx.x% | xx.x% | XX.X% | XX.X% | xx.x% |
| Failure | XX.X% | XX.X% | XX.X% | XX.X% | XX.X% | XX.X% |
| | | | | to 40 years | DTV 1702 | DTW 1502 |
| | W.1.:.1. OD | W.1.1.1. DID | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| > 2 C - 1 D - 1 - 1 - 1 - 1 - 1 | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | XX.X% | xx.x% | xx.x% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% |

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.4: Responder Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population - Responders)


| | Baseline Inflammatory Lesion Count < median (xx) | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | N=xx | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | | | | | | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | XX.X% | xx.x% | XX.X% | XX.X% | xx.x% | xx.x% |
| Failure | xx.x% | XX.X% | xx.x% | $XX.X^{0}/_{0}$ | xx.x% | $XX.X^{0}/_{0}$ |
| | | Baseli | • | Lesion Count≥ med | lian (xx) | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | | | | | | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | $XX.X^{0}/_{0}$ | $XX.X^{0}/_{0}$ | $XX.X^{0}/_{0}$ | $XX.X^{0}/_{0}$ | xx.x% | XX.X% |
| Failure | XX.X% | XX.X% | XX.X% | xx.x% | xx.x% | XX.X% |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.4: Responder Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population - Responders)


| | Baseline Non-Inflammatory Lesion Count < median (xx) | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | (N=xx) | N=xx | (N=xx) |
| >= 2 Grade Reduction from Baseline and | | | | | | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | $XX.X^{0}/_{0}$ |
| Failure | XX.X% | $XX.X^{0}/_{0}$ | XX.X% | $XX.X^{0}/_{0}$ | xx.x% | $XX.X^{0}/_{0}$ |
| | | Baseline | Non-Inflammator | y Lesion Count≥n | nedian (xx) | |
| | | Baseline | Non-Inflammator<br>Vehicle | y Lesion Count≥n<br>BTX 1503 | nedian (xx)<br>BTX 1503 | BTX 1503 |
| | Vehicle QD | <b>Baseline</b> Vehicle BID | | • | , , | BTX 1503<br>2.5% QD |
| | Vehicle QD (N=xx) | | Vehicle | BTX 1503 | BTX 1503 | |
| >= 2 Grade Reduction from Baseline and | | Vehicle BID | Vehicle<br>Combined | BTX 1503<br>5% BID | BTX 1503<br>5% QD | 2.5% QD |
| >= 2 Grade Reduction from Baseline and IGA Grade of 0 or 1 | | Vehicle BID | Vehicle<br>Combined | BTX 1503<br>5% BID | BTX 1503<br>5% QD | 2.5% QD |
| | | Vehicle BID (N=xx) xx.x% | Vehicle<br>Combined | BTX 1503<br>5% BID | BTX 1503<br>5% QD | 2.5% QD |
| IGA Grade of 0 or 1 | (N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | 2.5% QD<br>(N=xx) |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.4: Responder Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population - Responders)


| | Baseline Total Lesion Count < median (xx) | | | | | |
|---|---|---|---|---|---|---|
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | | | <del></del> _ | | <del></del> _ | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | XX.X% | XX.X% | xx.x% | XX.X% | XX.X% |
| Failure | XX.X% | xx.x% | XX.X% | XX.X% | xx.x% | $XX.X^{0}/_{0}$ |
| | | В | aseline Total Lesio | n Count ≥ median | (xx) | |
| | | В | aseline Total Lesio<br>Vehicle | n Count≥ median<br>BTX 1503 | ( <b>xx</b> )<br>BTX 1503 | BTX 1503 |
| | Vehicle QD | B<br>Vehicle BID | | | ` / | BTX 1503<br>2.5% QD |
| | Vehicle QD<br>(N=xx) | | Vehicle | BTX 1503 | BTX 1503 | |
| >= 2 Grade Reduction from Baseline and | | Vehicle BID | Vehicle<br>Combined | BTX 1503<br>5% BID | BTX 1503<br>5% QD | 2.5% QD |
| >= 2 Grade Reduction from Baseline and IGA Grade of 0 or 1 | | Vehicle BID | Vehicle<br>Combined | BTX 1503<br>5% BID | BTX 1503<br>5% QD | 2.5% QD |
| | | Vehicle BID | Vehicle<br>Combined | BTX 1503<br>5% BID | BTX 1503<br>5% QD | 2.5% QD |
| IGA Grade of 0 or 1 | (N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | 2.5% QD<br>(N=xx) |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.4: Responder Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population - Responders)


| | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Baseline IGA Vehicle Combined (N=xx) | of 3 (Moderate) BTX 1503 5% BID (N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| >= 2 Grade Reduction from Baseline and IGA Grade of 0 or 1 | | | | | | |
| Success | XX.X% | XX.X% | XX.X <sup>0</sup> / <sub>0</sub> | XX.X% | xx.x% | XX.X% |
| Failure | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% |
| | | | Baseline IG | A of 4 (Severe) | | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | N=xx | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and | | | | | | |
| IGA Grade of 0 or 1 | | | | | | |
| Success | XX.X% | xx.x% | XX.X% | XX.X% | XX.X% | XX.X% |
| Failure | XX.X% | XX.X% | XX.X <sup>0</sup> / <sub>0</sub> | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | XX.X% |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.2.3.4: Responder Subgroup Summary of Secondary Efficacy Endpoint: Dichotomized IGA at Day 84 (PP Population - Responders)


| | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Percent Complian Vehicle Combined (N=xx) | ce < median (xx.x%<br>BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| >= 2 Grade Reduction from Baseline and IGA Grade of 0 or 1 | | | | | | |
| Success<br>Failure | XX.X%<br>XX.X% | XX.X%<br>XX.X% | xx.x%<br>xx.x% | xx.x%<br>xx.x% | xx.x%<br>xx.x% | xx.x%<br>xx.x% |
| | | | Percent Complian | ce≥ median (xx.x% | (o) | |
| | | | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 |
| | Vehicle QD | Vehicle BID | Combined | 5% BID | 5% QD | 2.5% QD |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| >= 2 Grade Reduction from Baseline and IGA Grade of 0 or 1 | | | | | | |
| Success | xx.x% | XX.X% | $XX.X^{0}/_{0}$ | XX.X% | $XX.X^{0}/_{0}$ | xx.x% |
| Failure | XX.X% | XX.X% | XX.X% | XX.X% | XX.X% | XX.X% |

Note: Responder is defined as upper 80<sup>th</sup> percentile showing absolute reduction in inflammatory lesions from Baseline. No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.3.1.1: Exploratory Efficacy Endpoint: Summary of Inflammatory Lesion Count by Visit (ITT Population) (Page x of y)

| Baseline | Vehicle QD (N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | xx, xx | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx |

Note: Missing values imputed using LOCF.




Date: 24 MAY 2019

Table 14.2.3.1.1: Exploratory Efficacy Endpoint: Summary of Inflammatory Lesion Count by Visit (ITT Population)
(Page x of y)

| Day 14 | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Change from Baseline | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX,XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | xx, xx | xx, xx | XX, XX | XX, XX |
| Percent Change from Baseline | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

[Continue for Day 28, Day 56, and Day 84]

Note: Missing values imputed using LOCF.




Date: 24 MAY 2019

Repeat Table 14.2.3.1.1 for the following:

Table 14.2.3.1.2: Exploratory Efficacy Endpoint: Summary of Inflammatory Lesion Count by Visit (PP Population)

Programming note: replace last footnote with:

Note: No imputations were made for missing data.

Table 14.2.3.2.1: Exploratory Efficacy Endpoint: Summary of Non-Inflammatory Lesion Count by Visit (ITT Population)

Table 14.2.3.2.2: Exploratory Efficacy Endpoint: Summary of Non-Inflammatory Lesion Count by Visit (PP Population)

Programming note: replace last footnote with:

Note: No imputations were made for missing data.

Table 14.2.3.3.1: Exploratory Efficacy Endpoint: Summary of Total Lesion Count by Visit (ITT Population)

Table 14.2.3.3.2: Exploratory Efficacy Endpoint: Summary of Total Lesion Count by Visit (PP Population)

Programming note: replace last footnote with:

Note: No imputations were made for missing data.



Botanix BTX.2018.001

Version: v1 Date: 24 MAY 2019

Table 14.2.3.4.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Inflammatory Lesion Count at Day 84 (Comparing Dose Frequencies)

(ITT Population) 

| Change from Baseline in<br>Inflammatory Lesion Counts | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>QD Combined<br>(N=xx) |
|---|---|---|---|---|---|---|
| LSMean <sup>a</sup> | XX.X | XX.X | XX.X | XX.X | XX.X | |
| LSSD <sup>a</sup> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | |
| Unranked P-value vs. Vehicle <sup>a</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Vehicle <sup>b</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| LSMean <sup>c</sup> | XX.X | | | | | XX.X |
| LSSD <sup>c</sup> | XX.XX | | | | | XX.XX |
| Unranked P-value vs. Vehicle <sup>c</sup><br>Ranked P-value vs. Vehicle <sup>d</sup> | | | | | | 0.xxxx<br>0.xxxx |

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from an analysis of variance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>b</sup> Contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>c</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 QD combined compared to vehicle QD) from an analysis of variance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>d</sup> Contrast p-values (BTX 1503 QD combined compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion counts as the covariate.

Note: Missing values imputed using LOCF.



Botanix BTX.2018.001

Version: v1 Date: 24 MAY 2019

Table 14.2.3.4.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Inflammatory Lesion Count at Day 84 (Comparing

Dose Frequencies) (ITT Population) 

| Percent Change from Baseline in<br>Inflammatory Lesion Counts<br>LSMean <sup>a</sup><br>LSSD <sup>a</sup><br>Unranked P-value vs. Vehicle <sup>a</sup><br>Ranked P-value vs. Vehicle <sup>b</sup> | Vehicle QD (N=xx) xx.x xx.xx | Vehicle BID (N=xx) xx.x xx.xx | BTX 1503 5% BID (N=xx) xx.x xx.xx 0.xxxx 0.xxxx | BTX 1503 5% QD (N=xx) xx.x xx.xx 0.xxxx | BTX 1503 2.5% QD (N=xx) xx.x xx.xx 0.xxxx | BTX 1503<br>QD Combined<br>(N=xx) |
|---|---|---|---|---|---|---|
| LSMean <sup>c</sup><br>LSSD <sup>c</sup><br>Unranked P-value vs. Vehicle <sup>c</sup><br>Ranked P-value vs. Vehicle <sup>d</sup> | xx.x<br>xx.xx | | | | | xx.x<br>xx.xx<br>0.xxxx<br>0.xxxx |

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from an analysis of variance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>b</sup> Contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>c</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 QD combined compared to vehicle QD) from an analysis of variance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>d</sup> Contrast p-values (BTX 1503 QD combined compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion counts as the covariate.

Note: Missing values imputed using LOCF.




Date: 24 MAY 2019

Repeat Table 14.2.3.4.1 for the following:

Table 14.2.3.4.2: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Inflammatory Lesion Count at Day 84 (Comparing Dose Frequencies) (PP Population)

Programming note: replace last footnote with: Note: No imputations were made for missing data.

Table 14.2.3.5.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (Comparing Dose Frequencies) (ITT Population)

Table 14.2.3.5.2: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Non-Inflammatory Lesion Count at Day 84 (Comparing Dose Frequencies) (PP Population)

Programming note: replace last footnote with:

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.3.6.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Inflammatory Lesion Count by Visit (ITT Population)


| | Vehicle | BTX 1503 | BTX 1503 | BTX 1503 | C1 |
|---|---|---|---|---|---|
| | Combined | 5% BID | 5% QD | 2.5% QD | Skewness |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | P-value |
| Change from Baseline in | | | | | |
| Inflammatory Lesion Counts | | | | | |
| Day 14 | | | | | |
| LSMean <sup>a</sup> | XX.X | XX.X | XX.X | XX.X | $0.xxxx^b$ |
| $LSSD^a$ | XX.XX | XX.XX | XX.XX | XX.XX | |
| Unranked P-value vs. Combined Vehicle <sup>a</sup> | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Combined Vehicle <sup>c</sup> | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Day 28 | | | | | |
| LSMean <sup>a</sup> | XX.X | XX.X | XX.X | XX.X | $0.xxxx^b$ |
| LSSD <sup>a</sup> | XX.XX | XX.XX | XX.XX | XX.XX | |
| Unranked P-value vs. Combined Vehicle <sup>a</sup> | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Combined Vehicle <sup>c</sup> | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Day 56 | | | | | |
| LSMean <sup>a</sup> | XX.X | XX.X | XX.X | XX.X | $0.xxxx^b$ |
| LSSD <sup>a</sup> | XX.XX | XX,XX | XX.XX | XX.XX | |
| Unranked P-value vs. Combined Vehicle <sup>a</sup> | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Combined Vehicle <sup>c</sup> | | 0.xxxx | 0.xxxx | 0.xxxx | |

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values from an analysis of covariance with factors of treatment group (vehicle treatment groups included as single combined treatment group) and corresponding baseline lesion count as the covariate.

Note: Missing values imputed using LOCF.

<sup>&</sup>lt;sup>b</sup> Skewness test is based on methods presented by J.H. Zar (1984).

<sup>&</sup>lt;sup>c</sup> Contrast p-values from a ranked analysis of covariance with factors of treatment group (vehicle treatment groups included as single combined treatment group) and corresponding baseline lesion count as the covariate.




Date: 24 MAY 2019

Table 14.2.3.6.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Inflammatory Lesion Count by Visit (ITT Population)


| Percent Change from Baseline in | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | Skewness<br>P-value |
|---|---|---|---|---|---|
| Inflammatory Lesion Counts | | | | | |
| Day 14 | | | | | o h |
| LSMean <sup>a</sup> | XX.X | XX.X | XX.X | XX.X | $0.xxxx^b$ |
| LSSD <sup>a</sup> | XX.XX | XX.XX | XX.XX | XX.XX | |
| Unranked P-value vs. Combined Vehicle <sup>a</sup> | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Combined Vehicle <sup>c</sup> | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Day 28 | | | | | |
| LSMean <sup>a</sup> | XX.X | XX.X | XX.X | XX.X | $0.xxxx^b$ |
| $LSSD^a$ | XX.XX | XX.XX | XX.XX | XX.XX | |
| Unranked P-value vs. Combined Vehicle <sup>a</sup> | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Combined Vehicle <sup>c</sup> | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Day 56 | | | | | |
| LSMean <sup>a</sup> | XX.X | XX.X | XX.X | XX.X | $0.xxxx^b$ |
| LSSD <sup>a</sup> | XX.XX | XX.XX | XX.XX | XX.XX | |
| Unranked P-value vs. Combined Vehicle <sup>a</sup> | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Combined Vehicle <sup>c</sup> | | 0.xxxx | 0.xxxx | 0.xxxx | |

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values from an analysis of covariance with factors of treatment group (vehicle treatment groups included as single combined treatment group) and corresponding baseline lesion count as the covariate.

Note: Missing values imputed using LOCF.

<sup>&</sup>lt;sup>b</sup> Skewness test is based on methods presented by J.H. Zar (1984).

<sup>&</sup>lt;sup>c</sup> Contrast p-values from a ranked analysis of covariance with factors of treatment group (vehicle treatment groups included as single combined treatment group) and corresponding baseline lesion count as the covariate.




Date: 24 MAY 2019

Repeat Table 14.2.3.6.1 for the following:

Table 14.2.3.6.2: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Inflammatory Lesion Count by Visit (PP Population)

Programming note: replace last footnote with:

Note: No imputations were made for missing data.

Table 14.2.3.7.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Non-Inflammatory Lesion Count by Visit (ITT Population)

Table 14.2.3.7.2: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Non-Inflammatory Lesion Count by Visit (PP Population)

Programming note: replace last footnote with:

Note: No imputations were made for missing data.

Table 14.2.3.8.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Total Lesion Count by Visit (ITT Population)

Table 14.2.3.8.2: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Total Lesion Count by Visit (PP Population) *Programming note: replace last footnote with:* 

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.3.9.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Inflammatory Lesion Count by Visit (Comparing Dose Frequencies)

(ITT Population) 

| Change from Baseline in<br>Inflammatory Lesion Counts<br>Day 14 | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>QD Combined<br>(N=xx) |
|---|---|---|---|---|---|---|
| LSMean <sup>a</sup> | XX.X | XX.X | XX.X | XX.X | XX.X | |
| LSSD <sup>a</sup> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | |
| Unranked P-value vs. Vehicle <sup>a</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Vehicle <sup>b</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| LSMean <sup>c</sup> | XX.X | | | | | XX.X |
| $LSSD^{c}$ | XX.XX | | | | | XX.XX |
| Unranked P-value vs. Vehicle <sup>c</sup> | | | | | | 0.xxxx |
| Ranked P-value vs. Vehicled | | | | | | 0.xxxx |

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from an analysis of variance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>b</sup> Contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>c</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 QD combined compared to vehicle QD) from an analysis of variance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>d</sup> Contrast p-values (BTX 1503 QD combined compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion counts as the covariate.

Note: Missing values imputed using LOCF.




Date: 24 MAY 2019

Table 14.2.3.9.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Inflammatory Lesion Count by Visit (Comparing Dose Frequencies)

(ITT Population) 

| Change from Baseline in<br>Inflammatory Lesion Counts<br>Day 28 | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>QD Combined<br>(N=xx) |
|---|---|---|---|---|---|---|
| LSMean <sup>a</sup> | XX.X | XX.X | XX.X | XX.X | XX.X | |
| LSSD <sup>a</sup> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | |
| Unranked P-value vs. Vehicle <sup>a</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Vehicle <sup>b</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| LSMean <sup>c</sup> | XX.X | | | | | XX.X |
| $LSSD^{c}$ | XX.XX | | | | | XX.XX |
| Unranked P-value vs. Vehicle <sup>c</sup> | | | | | | 0.xxxx |
| Ranked P-value vs. Vehicle <sup>d</sup> | | | | | | 0.xxxx |

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from an analysis of variance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

#### SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>b</sup> Contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>c</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 QD combined compared to vehicle QD) from an analysis of variance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>d</sup> Contrast p-values (BTX 1503 QD combined compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion counts as the covariate.

Note: Missing values imputed using LOCF.




Date: 24 MAY 2019

Table 14.2.3.9.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Inflammatory Lesion Count by Visit (Comparing Dose Frequencies)

(ITT Population) 

| Change from Baseline in<br>Inflammatory Lesion Counts<br>Day 56 | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>QD Combined<br>(N=xx) |
|---|---|---|---|---|---|---|
| LSMean <sup>a</sup> | XX.X | XX.X | XX.X | XX.X | XX.X | |
| LSSD <sup>a</sup> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | |
| Unranked P-value vs. Vehicle <sup>a</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Vehicle <sup>b</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| LSMean <sup>c</sup> | XX.X | | | | | XX.X |
| $LSSD^{c}$ | XX.XX | | | | | XX.XX |
| Unranked P-value vs. Vehicle <sup>c</sup> | | | | | | 0.xxxx |
| Ranked P-value vs. Vehicle <sup>d</sup> | | | | | | 0.xxxx |

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from an analysis of variance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

#### SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>b</sup> Contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>c</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 QD combined compared to vehicle QD) from an analysis of variance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>d</sup> Contrast p-values (BTX 1503 QD combined compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion counts as the covariate.

Note: Missing values imputed using LOCF.




Date: 24 MAY 2019

Table 14.2.3.9.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Inflammatory Lesion Count by Visit (Comparing Dose Frequencies)

(ITT Population) 

| Percent Change from Baseline in<br>Inflammatory Lesion Counts<br>Day 14 | Vehicle QD (N=xx) | Vehicle BID (N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>QD Combined<br>(N=xx) |
|---|---|---|---|---|---|---|
| LSMean <sup>a</sup> | XX.X | XX.X | XX.X | XX.X | XX.X | |
| LSSD <sup>a</sup> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | |
| Unranked P-value vs. Vehicle <sup>a</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Vehicle <sup>b</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| LSMean <sup>c</sup> | XX.X | | | | | XX.X |
| LSSD <sup>c</sup> | XX.XX | | | | | XX.XX |
| Unranked P-value vs. Vehicle <sup>c</sup> | | | | | | 0.xxxx |
| Ranked P-value vs. Vehicle <sup>d</sup> | | | | | | 0.xxxx |

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from an analysis of variance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

#### SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>b</sup> Contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>c</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 QD combined compared to vehicle QD) from an analysis of variance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion count as the covariate.

d Contrast p-values (BTX 1503 QD combined compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion counts as the covariate.

Note: Missing values imputed using LOCF.




Date: 24 MAY 2019

Table 14.2.3.9.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Inflammatory Lesion Count by Visit (Comparing Dose Frequencies)

(ITT Population) 

| Percent Change from Baseline in<br>Inflammatory Lesion Counts<br>Day 28 | Vehicle QD (N=xx) | Vehicle BID (N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>QD Combined<br>(N=xx) |
|---|---|---|---|---|---|---|
| LSMean <sup>a</sup> | XX.X | XX.X | XX.X | XX.X | XX.X | |
| LSSD <sup>a</sup> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | |
| Unranked P-value vs. Vehicle <sup>a</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Vehicle <sup>b</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| LSMean <sup>c</sup> | XX.X | | | | | XX.X |
| $LSSD^{c}$ | XX.XX | | | | | XX.XX |
| Unranked P-value vs. Vehicle <sup>c</sup> | | | | | | 0.xxxx |
| Ranked P-value vs. Vehicle <sup>d</sup> | | | | | | 0.xxxx |

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from an analysis of variance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

#### SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>b</sup> Contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>c</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 QD combined compared to vehicle QD) from an analysis of variance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>d</sup> Contrast p-values (BTX 1503 QD combined compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion counts as the covariate.

Note: Missing values imputed using LOCF.



Botanix BTX.2018.001

Version: v1 Date: 24 MAY 2019

Table 14.2.3.9.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Inflammatory Lesion Count by Visit (Comparing Dose Frequencies)

(ITT Population) 

| Percent Change from Baseline in<br>Inflammatory Lesion Counts<br>Day 56 | Vehicle QD (N=xx) | Vehicle BID (N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>QD Combined<br>(N=xx) |
|---|---|---|---|---|---|---|
| LSMean <sup>a</sup> | XX.X | XX.X | XX.X | XX.X | XX.X | |
| LSSD <sup>a</sup> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | |
| Unranked P-value vs. Vehicle <sup>a</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| Ranked P-value vs. Vehicle <sup>b</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| LSMean <sup>c</sup> | XX.X | | | | | XX.X |
| LSSD <sup>c</sup> | XX.XX | | | | | XX.XX |
| Unranked P-value vs. Vehicle <sup>c</sup> | | | | | | 0.xxxx |
| Ranked P-value vs. Vehicle <sup>d</sup> | | | | | | 0.xxxx |

<sup>&</sup>lt;sup>a</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from an analysis of variance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

#### SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>b</sup> Contrast p-values (BTX 1503 BID group compared to vehicle BID and each BTX 1503 QD group compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (no treatment groups combined) and corresponding baseline lesion count as the covariate.

<sup>&</sup>lt;sup>c</sup> Least squares mean, standard deviation, and contrast p-values (BTX 1503 QD combined compared to vehicle QD) from an analysis of variance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion count as the covariate.

d Contrast p-values (BTX 1503 QD combined compared to vehicle QD) from a ranked analysis of covariance with factors of treatment group (BTX 1503 QD treatment groups combined) and corresponding baseline lesion counts as the covariate.

Note: Missing values imputed using LOCF.




Date: 24 MAY 2019

Repeat Table 14.2.3.9.1 for the following:

Table 14.2.3.9.2: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Inflammatory Lesion Count by Visit (Comparing Dose Frequencies) (PP Population)

Programming note: replace last footnote with: Note: No imputations were made for missing data.

Table 14.2.3.10.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Non-Inflammatory Lesion Count by Visit (Comparing Dose Frequencies) (ITT Population)

Table 14.2.3.10.2: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Non-Inflammatory Lesion Count by Visit (Comparing Dose Frequencies) (PP Population)

Programming note: replace last footnote with:

Note: No imputations were made for missing data.

Table 14.2.3.11.1: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Total Lesion Count by Visit (Comparing Dose Frequencies) (ITT Population)

Table 14.2.3.11.2: Exploratory Efficacy Endpoint: Analysis of Absolute and Percent Change from Baseline in Total Lesion Count by Visit (Comparing Dose Frequencies) (PP Population)

Programming note: replace last footnote with: Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.3.12.1: Exploratory Efficacy Endpoint: Summary of IGA Score by Visit (ITT Population)

| Baseline | Vehicle QD<br>(N=xx) | Vehicle BID<br>_(N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX |
| 0 Clear | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) |
| 2 Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) |
| 3 Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX,X |
| Min., Max. | XX, XX | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx |

[Repeat for Day 14, Day 28, Day 56, and Day 84]

Note: Missing values imputed using LOCF.




Date: 24 MAY 2019

Repeat Table 14.2.3.12.1 for the following:

Table 14.2.3.12.2: Exploratory Efficacy Endpoint: Summary of IGA Score by Visit (PP Population)

Programming note: replace last footnote with: Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.3.13.1: Exploratory Efficacy Endpoint: Analysis of Dichotomized IGA at Day 84 (Comparing Dose Frequencies) (ITT Population)

| >= 2 Grade Reduction from Baseline in IGA Success Failure P-value vs. Vehicle <sup>a</sup> P-value vs. Vehicle <sup>b</sup> | Vehicle QD<br>(N=xx)<br>xx.x%<br>xx.x% | Vehicle BID (N=xx) xx.x% xx.x% | BTX 1503<br>5% BID<br>(N=xx)<br>xx.x%<br>xx.x%<br>0.xxxx | BTX 1503<br>5% QD<br>(N=xx)<br>xx.x%<br>xx.x%<br>0.xxxx | BTX 1503<br>2.5% QD<br>(N=xx)<br>xx.x%<br>xx.x%<br>0.xxxx | BTX 1503 QD Combined (N=xx) xx.x% xx.x% 0.xxxx | Treatment P-value 0.xxxxa |
|---|---|---|---|---|---|---|---|
| IGA Grade of 0 or 1 Success Failuire P-value vs. Vehicle <sup>a</sup> P-value vs. Vehicle <sup>b</sup> | xx.x%<br>xx.x% | xx.x%<br>xx.x% | xx.x%<br>xx.x%<br>0.xxxx | xx.x%<br>xx.x%<br>0.xxxx | xx.x%<br>xx.x%<br>0.xxxx | xx.x%<br>xx.x%<br>0.xxxx | 0.xxxx <sup>a</sup> |
| >= 2 Grade Reduction from Baseline and IGA Grade of 0 or 1 Success Failure P-value vs. Vehicle <sup>a</sup> P-value vs. Vehicle <sup>b</sup> | xx.x%<br>xx.x% | xx.x%<br>xx.x% | xx.x%<br>xx.x%<br>0.xxxx | xx.x%<br>xx.x%<br>0.xxxx | xx.x%<br>xx.x%<br>0.xxxx | xx.x%<br>xx.x%<br>0.xxxx | 0.xxxx <sup>a</sup> |

<sup>&</sup>lt;sup>a</sup> P-value from a logistic regression with factor of treatment group (no treatment groups combined) where BTX 1503 BID group is compared to vehicle BID and each BTX 1503 QD group is compared to vehicle QD.

Note: Missing values imputed using LOCF.

<sup>&</sup>lt;sup>b</sup> P-value from a logistic regression with factor of treatment group (BTX 1503 QD treatment groups combined) where BTX 1503 combined QD group is compared to vehicle QD.




Date: 24 MAY 2019

Repeat Table 14.2.3.13.1 for the following:

Table 14.2.3.13.2: Exploratory Efficacy Endpoint: Analysis of Dichotomized IGA at Day 84 (Comparing Dose Frequencies) (PP Population)

Programming note: replace last footnote with:

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.3.14.1: Exploratory Efficacy Endpoint: Analysis of Dichotomized IGA by Visit (ITT Population)

| Day 14 | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | Treatment P-value |
|---|---|---|---|---|---|---|---|
| >= 2 Grade Reduction from Baseline in IGA | | | | | | | $0.xxxx^a$ |
| Success | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | ********* |
| Failure | xx.x% | XX.X% | XX.X% | xx.x% | XX.X% | XX.X% | |
| P-value vs. Combined Vehicle <sup>a</sup> | | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| IGA Grade of 0 or 1 | | | | | | | $0.xxxx^a$ |
| Success | xx.x% | xx.x% | XX.X% | XX.X% | $XX.X^{0}/_{0}$ | xx.x% | |
| Failure | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | |
| P-value vs. Combined Vehicle <sup>a</sup> | | | | 0.xxxx | 0.xxxx | 0.xxxx | |
| >= 2 Grade Reduction from Baseline and IGA<br>Grade of 0 or 1 | | | | | | | 0.xxxx <sup>a</sup> |
| Success | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | XX.X% | |
| Failure | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | |
| P-value vs. Combined Vehicle <sup>a</sup> | | | | 0.xxxx | 0.xxxx | 0.xxxx | |

[repeat for Day 28 and Day 56]

<sup>&</sup>lt;sup>a</sup> P-value from a logistic regression with factor of treatment group (vehicle treatment groups included as single combined treatment group). Note: Missing values imputed using LOCF.




Date: 24 MAY 2019

Repeat Table 14.2.3.14.1 for the following:

Table 14.2.3.14.2: Exploratory Efficacy Endpoint: Analysis of Dichotomized IGA by Visit (PP Population)

Programming note: replace last footnote with: Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.3.15.1: Exploratory Efficacy Endpoint: Analysis of Dichotomized IGA by Visit (Comparing Dose Frequencies) (ITT Population)

| | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>QD Combined<br>(N=xx) | Treatment P-value |
|---|---|---|---|---|---|---|---|
| Day 14 | | | | | | | 0 3 |
| >= 2 Grade Reduction from Baseline in IGA | | 0/ | 0/ | 0/ | 0/ | 0/ | $0.xxxx^a$ |
| Success | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | |
| Failure | XX.X% | XX.X% | xx.x% | xx.x% | XX.X% | xx.x% | |
| P-value vs. Vehicle <sup>a</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | | |
| P-value vs. Vehicle <sup>b</sup> | | | | | | 0.xxxx | |
| IGA Grade of 0 or 1 | | | | | | | 0.xxxx <sup>a</sup> |
| Success | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | |
| Failuire | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | |
| P-value vs. Vehicle <sup>a</sup> | 7171.717 | 7171.7170 | 0.xxxx | 0.xxxx | 0.xxxx | 717.717 0 | |
| P-value vs. Vehicle <sup>b</sup> | | | U.AAAA | U.AAAA | U.AAAA | 0 **** | |
| r-value vs. Vehicle | | | | | | 0.xxxx | |
| >= 2 Grade Reduction from Baseline and | | | | | | | $0.xxxx^a$ |
| IGA Grade of 0 or 1 | | | | | | | |
| Success | xx.x% | xx.x% | xx.x% | XX.X% | xx.x% | xx.x% | |
| Failure | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | |
| P-value vs. Vehicle <sup>a</sup> | | | 0.xxxx | 0.xxxx | 0.xxxx | | |
| P-value vs. Vehicle <sup>b</sup> | | | VIIII | O.IIIIII | omi | 0.xxxx | |
| [variet for Day 28 and Day 56] | | | | | | V.MAA | |

[repeat for Day 28 and Day 56]

Note: Missing values imputed using LOCF.

<sup>&</sup>lt;sup>a</sup> P-value from a logistic regression with factor of treatment group (no treatment groups combined) where BTX 1503 BID group is compared to vehicle BID and each BTX 1503 QD group is compared to vehicle QD.

<sup>&</sup>lt;sup>b</sup> P-value from a logistic regression with factor of treatment group (BTX 1503 QD treatment groups combined) where BTX 1503 combined QD group is compared to vehicle QD.




Date: 24 MAY 2019

Repeat Table 14.2.3.15.1 for the following:

Table 14.2.3.15.2: Exploratory Efficacy Endpoint: Analysis of Dichotomized IGA by Visit (Comparing Dose Frequencies) (PP Population)

Programming note: replace last footnote with:

Note: No imputations were made for missing data.




Date: 24 MAY 2019

Table 14.2.3.16.1: Exploratory Efficacy Endpoint: Summary of Acne Patient Self-Questionnaire (ITT Population)

| Z.16 Donordion | Vehicle QD (N=xx) | Vehicle BID<br>(N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| Self-Perception<br>Baseline | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 84 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx | XX, XX |
| Change from Baseline | | | | | | |
| n | xx | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

[Repeat for Role-Social, Role-Emotional, and Acne Symptoms]




Date: 24 MAY 2019

Repeat Table 14.2.3.16.1 for the following:

Table 14.2.3.16.2: Exploratory Efficacy Endpoint: Summary of Acne Patient Self-Questionnaire (PP Population)




Date: 24 MAY 2019

Table 14.2.3.17.1: Exploratory Efficacy Endpoint: Summary of Patient Reported Outcome (ITT Population)

| | Vehicle QD<br>(N=xx) | Vehicle BID<br>(N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|---|
| Compared to the beginning of treatment, my acne is: | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Much Better | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Slightly Better | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) |
| The Same | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Slightly Worse | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Much Worse | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |




Date: 24 MAY 2019

Repeat Table 14.2.3.17.1 for the following:

Table 14.2.3.17.2: Exploratory Efficacy Endpoint: Summary of Patient Reported Outcome (PP Population)




Date: 24 MAY 2019

Table 14.3.0.1: Summary of Extent of Exposure (Safety Population) 

| | Vehicle QD<br>(N=xx) | Vehicle BID<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|
| Exposure (Days) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | xx, xx | xx, xx | XX, XX | XX, XX | xx, xx |
| Amount of Study Drug Used Total (g) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | xx, xx | xx, xx | XX, XX | xx, xx | XX, XX |
| Average Amount of Study Drug Used Per Day (g/day) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | xx, xx | XX, XX | xx, xx | XX, XX | xx, xx |

<sup>&</sup>lt;sup>a</sup> Compliant with the dosing regimen is if the subject applied at least 80% but no more than 120% of expected applications while enrolled in the study. <sup>b</sup> Percentages based on the number of subjects in the safety population with percent compliance calculated.




Date: 24 MAY 2019

Table 14.3.0.1: Summary of Extent of Exposure (Safety Population) 

| | Vehicle QD<br>(N=xx) | Vehicle BID<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) |
|---|---|---|---|---|---|
| Number of Applications | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| Number of Missed Applications | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| Percent Compliance | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| Compliant <sup>a</sup> | | | | | |
| Yes <sup>b</sup> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No <sup>b</sup> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Compliant with the dosing regimen is if the subject applied at least 80% but no more than 120% of expected applications while enrolled in the study.

<sup>&</sup>lt;sup>b</sup> Percentages based on the number of subjects in the safety population with percent compliance calculated. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Table 14.3.0.2.1: Summary of Cutaneous Tolerability Assessments (Safety Population)
(Page x of y)

| Burning/Stinging Baseline | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>Combined<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX | XX |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| None | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Day 1 – 15 Mins Post-Dose | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Severe | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) | xx(xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Day 14 – Pre-Dose | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderare | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | , , | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| [Repeat for Day 14 – 15 Mins Post-I | , | ( ) | , , | , , | , | , | , |

[Repeat for Pruritus, Erythema, Dryness, and Scaling]

Note: Percentages are based on the number of subjects in each treatment group in the Safety population with a non-missing assessment at the given visit. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)




Date: 24 MAY 2019

Table 14.3.0.2.2: Summary of Cutaneous Tolerability Assessments Worst Post-Baseline Grades (Safety Population)
(Page x of y)

| Worst Post-Baseline Grade Burning/Stinging | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>Combined<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX | XX |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pruritus | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Erythema | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

[Repeat for Dryness and Scaling]

Note: Percentages are based on the number of subjects in each treatment group in the Safety population with at least one post-baseline assessment for the given category.




Date: 24 MAY 2019

Table 14.3.0.2.3: Summary of Mild, Moderate, or Severe Post-Baseline Cutaneous Tolerability Assessments (Safety Population)
(Page x of y)

| D (D I | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>Combined<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Post-Baseline | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Burning/Stinging | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pruritus | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Erythema | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Dryness | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Scaling | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Percentages are based on the number of subjects in each treatment group in the Safety population with at least one post-baseline assessment.




Date: 24 MAY 2019

Table 14.3.1.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population)

| Number (%) of Subjects Reporting At Least One<br>Treatment-Emergent Adverse Event<br>Number of Treatment-Emergent Adverse Events | Vehicle QD (N=xx) xx (xx.x%) | Vehicle BID (N=xx) xx (xx.x%) | Vehicle<br>Combined<br>(N=xx)<br>xx (xx.x%) | BTX 1503<br>5% BID<br>(N=xx)<br>xx ( xx.x%) | BTX 1503<br>5% QD<br>(N=xx)<br>xx ( xx.x%) | BTX 1503<br>2.5% QD<br>(N=xx)<br>xx ( xx.x%) | BTX 1503<br>Combined<br>(N=xx)<br>xx (xx.x%) |
|---|---|---|---|---|---|---|---|
| Number (%) of Subjects Reporting At Least One Serious<br>Treatment-Emergent Adverse Event<br>Number of Serious Treatment-Emergent Adverse Events | xx ( xx.x%) | | xx ( xx.x%) | | xx ( xx.x%) | | xx ( xx.x%) |
| Number (%) of Subjects who Discontinued Study Due to At Least One Treatment-Emergent Event Number of Treatment-Emergent Adverse Events Leading | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | xx | xx | xx | xx | xx | xx | xx |
| to Discontinuation of Study Maximum Severity Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate Mild Strongest Relationship to Study Drug | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Related | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Related | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the date of first application of study drug. Percentages are based on the number of subjects in each treatment group in the Safety population.

Related adverse events include possibly, probably, and definitely responses to relationship to study drug question.




Date: 24 MAY 2019

Table 14.3.1.1.2: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)

| System Organ Class <sup>a</sup><br>Preferred Term | Vehicle QD<br>(N=xx) | Vehicle BID (N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>Combined<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| System Organ Class 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | ` / | ` / | ` / | xx ( xx.x%) | , | ` / | ` / |
| Preferred Term x | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

. . .

Note: MedDRA Version 20.0.

Treatment-emergent adverse events are those with an onset on or after the date of first application of study drug.

Percentages are based on the number of subjects in each treatment group in the Safety population.

<sup>&</sup>lt;sup>a</sup> At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.




Repeat Table 14.3.1.1.2 for the following:

Table 14.3.1.1.3: Summary of Serious Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)

Table 14.3.1.1.4: Summary of Related Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population) Programming note: Add footnote –

Related adverse events include possibly, probably, and definitely responses to relationship to study drug question.

Table 14.3.1.1.5: Summary of Severe Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)

Table 14.3.1.1.6: Summary of Treatment-Emergent Adverse Events Leading to Study Discontinuation by MedDRA System Organ Class and Preferred Term (Safety Population)

Table 14.3.1.1.7: Summary of Treatment-Emergent Abuse-Related Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)




Table 14.3.1.2.1.1: Summary of Chemistry Results by Visit (Safety Population)

| Test Name (Units) Baseline | Vehicle QD<br>(N=xx) | Vehicle BID<br>(N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>Combined<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 84 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Change from Baseline | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min., Max. | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |

[repeat for each test]

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Programming note: Chemistry tests include: Glucose, Albumin, Total Protein, Calcium, Sodium, Potassium, Chloride, CO<sub>2</sub> (bicarbonate), BUN, Creatinine, Alkaline Phosphatase, ALT, AST, and Total Bilirubin. Test names will be standardized to CDISC Controlled Terminology.




Date: 24 MAY 2019

Table 14.3.1.2.1.2: Shift Table for Chemistry Results (Safety Population)

| Test Name (Units) | | _ | Baseline (N=xx) | |
|---|---|---|---|---|
| Vehicle QD (N=xx) | Day 84 (Na=xx) | BNL | WNL | ANL |
| | BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | ANL | xx (xx.x%) | xx(xx.x%) | xx ( xx.x%) |
| Vehicle BID (N=xx) | Day 84 (N <sup>a</sup> =xx) | | | |
| , | BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Vehicle Combined (N=xx) | Day 84 (Na=xx) | | | |
| , , | BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | ANL | xx ( xx.x%) | xx ( xx.x%) | xx(xx.x%) |

Note: BNL=Below Normal Limit, WNL=Within Normal Limit, ANL=Above Normal Limit.

Percentages are based on the number of subjects in the Safety population with both Baseline and Day 84 results.

<sup>&</sup>lt;sup>a</sup> Number of subjects with both Baseline and Day 84 results for the given treatment group.




Date: 24 MAY 2019

Table 14.3.1.2.1.2: Shift Table for Chemistry Results (Safety Population)

| Test Name (Units) | | | Baseline | |
|---|---|---|---|---|
| BTX 1503 5% BID (N=xx) | Day 84 ( $N^a=xx$ ) | BNL | WNL | ANL |
| ` , | BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| BTX 1503 5% QD (N=xx) | Day 84 (N <sup>a</sup> =xx) | | | |
| - , , | BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| BTX 1503 2.5% QD (N=xx) | Day 84 (Na=xx) | | | |
| | BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| BTX 1503 Combined (N=xx) | Day 84 (Na=xx) | | | |
| , , | BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| [Repeat for all tests] | | | | |

<sup>&</sup>lt;sup>a</sup> Number of subjects with both Baseline and Day 84 results for the given treatment group.

Note: BNL=Below Normal Limit, WNL=Within Normal Limit, ANL=Above Normal Limit.

Percentages are based on the number of subjects in the Safety population with both Baseline and Day 84 results.




Date: 24 MAY 2019

Repeat Table 14.3.1.2.1.1 for the following:

Table 14.3.1.2.2.1: Summary of CBC Results by Visit (Safety Population)

Programming note: CBC tests include: WBC (with differentials for ANC, Lymphocytes, monocytes, eosinophils, and basophils), RBC, Hemaglobin, Hematocrit, MCV, MCH, MCHC, and Platelet Count. Test names will be standardized to CDISC Controlled Terminology.

Repeat Table 14.3.1.2.1.2 for the following:

Table 14.3.1.2.2.2: Shift Table for CBC Results (Safety Population)

Repeat Table 14.3.1.2.1.1 for the following:

Table 14.3.1.2.3.1: Summary of Numeric Urinalysis Results by Visit (Safety Population)

Repeat Table 14.3.1.2.1.2 for the following:

Table 14.3.1.2.3.2: Shift Table for Numeric Urinalysis Results (Safety Population)




Date: 24 MAY 2019

Table 14.3.1.2.3.3: Summary of Character Urinalysis Results by Visit (Safety Population)

| Test Name (Units) Baseline | Vehicle QD<br>(N=xx) | Vehicle BID<br>(N=xx) | Vehicle<br>Combined<br>(N=xx) | BTX 1503<br>5% BID<br>(N=xx) | BTX 1503<br>5% QD<br>(N=xx) | BTX 1503<br>2.5% QD<br>(N=xx) | BTX 1503<br>Combined<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| n | XX | XX | XX | XX | XX | XX | XX |
| XXXXXXX | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| XXXXXXX | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| xxxxxxx | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Day 84 | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| XXXXXXX | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| XXXXXXX | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| XXXXXXX | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

[repeat for each test]

Note: Percentages are based on the number of subjects in the Safety population with a non-missing result for the given test and visit.



### Statistical Analysis Plan Botanix BTX.2018.001


Date: 24 MAY 2019

#### 11. INDEX OF PLANNED LISTINGS

| Listing 16.1.7: Randomization Scheme | 158 |
|---|---|
| Listing 16.2.1.1: Subject Disposition Information. | 159 |
| Listing 16.2.1.2: Discontinued Subjects | 160 |
| Listing 16.2.1.3: Screen Failures | 161 |
| Listing 16.2.2: Inclusion/Exclusion Criteria Not Met | 162 |
| Listing 16.2.3: Analysis Populations | 163 |
| Listing 16.2.4.1: Subject Demographic Information | 164 |
| Listing 16.2.4.2.1: Unique Medical History Coded to MedDRA System O | Organ Classes and Preferred Terms 165 |
| Listing 16.2.4.2.2: Medical History | 166 |
| Listing 16.2.4.2.3: Substance Use History | 167 |
| Listing 16.2.4.4.1: Unique Medication/Therapy Names Coded to WHO-D | DDE ATC Level 2 Terms and Preferred Names 168 |
| Listing 16.2.4.4.2: Prior and Concomitant Medications/Therapies | 169 |
| Listing 16.2.4.4.3: Unique Antibiotic Therapy Names Coded to WHO-DE | DE ATC Level 2 Terms and Preferred Names 170 |
| Listing 16.2.4.4.4: Concomitant Antibiotic Therapies | 171 |
| Listing 16.2.4.6: Physical Examination | 172 |
| Listing 16.2.5.1: Study Drug Administration | 173 |
| Listing 16.2.5.3: Drug Accountability | 174 |
| Listing 16.2.5.4: Dosing Compliance | 175 |
| Listing 16.2.5.5: Dosing Deviations | 176 |
| Listing 16.2.6.1: Lesion Count Evaluations | 177 |



### Statistical Analysis Plan Botanix BTX.2018.001


Date: 24 MAY 2019

| Listing 16.2.6.2: Investigator Global Assessment | 178 |
|---|---|
| Listing 16.2.6.3: Patient Reported Outcome Assessment | 179 |
| Listing 16.2.6.4: Acne-QoL Questionnaire. | 180 |
| Listing 16.2.6.5: Photography Information. | 181 |
| Listing 16.2.7.1: Cutaneous Tolerability Assessment | 182 |
| Listing 16.2.7.2.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Programme Coded to MedDRA System Organ Classes and Program Classes and | referred Terms 183 |
| Listing 16.2.7.2.2: Treatment-Emergent Adverse Events | 184 |
| Listing 16.2.7.2.3: Serious Adverse Events | 185 |
| Listing 16.2.7.2.4: Subjects Who Permanently Discontinued Study Drug and/or Discontinued | • |
| Listing 16.2.7.2.5: Unique Abuse-Related Adverse Events Coded to MedDRA System Organ | n Classes and Preferred Terms 187 |
| Listing 16.2.7.2.6: Treatment-Emergent Abuse-Related Adverse Events | 188 |
| Listing 16.2.8.1: Urine Pregnancy Test Results | 189 |
| Listing 16.2.8.2: Urine Drug Screen Results | 190 |
| Listing 16.2.8.2.1.1: Complete Blood Count Laboratory Test Results | 191 |
| Listing 16.2.8.2.1.2: Chemistry Laboratory Test Results | 192 |
| Listing 16.2.8.2.1.3: Urinalysis Laboratory Test Results | 192 |




Date: 24 MAY 2019

### Listing 16.1.7: Randomization Scheme (Page xx of yy)

| Subject | Age/Sex | Evaluable | Randomization<br>Number | Randomization<br>Date | Assigned<br>Treatment Group | Kit Dispensed<br>at Baseline |
|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxx | xxxx-xx-xx | xxxxxx xxxxxx xxxx | xxxxx |
| xxxxxx | XXXX | xxxxxxxx | xxxx | xxxx-xx-xx | xxxxxx | xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxx | xxxx-xx-xx | xxxxxx xxxxxx xxxx | XXXXX |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject.




Date: 24 MAY 2019

### Listing 16.2.1.1: Subject Disposition Information Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Evaluable | F: Date of First Dose L: Date (Day) 1 of Last Dose | Completion<br>Status | E: Date (Day) of Completion/Discontinuation R: Reason for Study Discontinuation | Additional Information <sup>2</sup> |
|---|---|---|---|---|
| S: xxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxx-xx-xx<br>L: xxxx-xx-xx (xx) | ****** | E: xxxx-xx-xx (xx) R: xxxxxx xxxxxxx xxxxxx | Cause of Death: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxx-xx-xx<br>L: xxxx-xx-xx (xx) | xxxxxxxx | E: xxxx-xx-xx (xx) R: xxxxxxxxx xx xxxxxxxx | |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxx-xx-xx<br>L: xxxx-xx-xx (xx) | XXXXXXXX | E: xxxx-xx-xx (xx)<br>R: xxxxxxxxx xx xxxxxxxx | |
| S: XXXXX<br>A: XXXX<br>E: XXXXXXXX | F: xxxx-xx-xx<br>L: xxxx-xx-xx (xx) | **** | E: xxxx-xx-xx (xx) R: xxxxxx xxxxxxx xxxxxx | Cause of Death: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>&</sup>lt;sup>2</sup> Additional information is collected on a conditional basis, all information collected is included in the listing. Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)




Date: 24 MAY 2019

### Listing 16.2.1.2: Discontinued Subjects Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Evaluable | F: Date of First Dose L: Date (Day) 1 of Last Dose | Completion<br>Status | E: Date (Day) 1 of<br>Completion/Discontinuation<br>R: Reason for Study<br>Discontinuation | Additional Information <sup>2</sup> |
|---|---|---|---|---|
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxx-xx-xx<br>L: xxxx-xx-xx (xx) | xxxxx xxxxxxxxx | E: xxxx-xx-xx (xx) R: xxxxxx xxxxxxx | Cause of Death: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxx-xx-xx<br>L: xxxx-xx-xx (xx) | xxxxxxxx | E: xxxx-xx-xx (xx)<br>R: xxxxxxxxxx xx xxxxxxxx | |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxx-xx-xx<br>L: xxxx-xx-xx (xx) | xxxxxxxx | E: xxxx-xx-xx (xx) R: xxxxxxxxxx xx xxxxxxxx | |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxxx | F: xxxx-xx-xx<br>L: xxxx-xx-xx (xx) | xxxxx xxxxxxxxxx | E: xxxx-xx-xx (xx) R: xxxxxx xxxxxxx xxxxxx | Cause of Death: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>2</sup> Additional information is collected on a conditional basis, all information collected is included in the listing.
Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



### Statistical Analysis Plan Botanix BTX.2018.001


Date: 24 MAY 2019

#### Listing 16.2.1.3: Screen Failures (Page x of xx)

| Subject | Age/Sex | Date of<br>Screen Failure | Reason for<br>Screen Failure |
|---|---|---|---|
| xxxxxxxx | xxxx | xxxx-xx-xx | xxxxxxxx xx xxxxxxx |
| xxxxxxxx | XXXX | xxxx-xx-xx | xxxx xx xxxxxx xx |
| xxxxxxxx | xxxx | xxxx-xx-xx | xxxxxxx xxxxx |




Date: 24 MAY 2019

## Listing 16.2.2: Inclusion/Exclusion Criteria Not Met Treatment Group (Page xx of yy)

| S: Subject A: Age/Sex E: Evaluable | V: Study Visit<br>D: Date | Inclusion/Exclusion<br>Criteria not met | Reason eligibility criteria not met |
|---|---|---|---|
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | V: xxxxxxxxxx<br>D: xxxx-xx-xx | xxxxxx<br>xxxxxx | XXXXX XXX XX XXXXXXXX XXXX XXXXXXXXXXX |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | V: xxxxxxxxxx<br>D: xxxx-xx-xx | xxxxxx | xxxxx xxx xx xxxxxxx xxxx xxxxxxxxxxxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | V: xxxxxxxxxx<br>D: xxxx-xx-xx | xxxxxx | ***** *** ** ******* **** ************ |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population.

Note: ITT = Intent-to-Treat Population; S = Salety Population; PP = Per-Protocol Population. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject and Criterion Failed.




Date: 24 MAY 2019

# Listing 16.2.3: Analysis Populations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Population | Included | Reason(s) Excluded |
|---|---|---|---|---|
| xxxxx | xxxx | Intent-to-Treat<br>Safety<br>Per-Protocol | xxx<br>xx | xxxxxxxxxx xxxxxxx xxxxxxxxxxxxxxxxxxx |
| xxxxx | XXXX | Intent-to-Treat<br>Safety<br>Per-Protocol | xxx<br>xxx<br>xx | ************ ************************* |
| xxxxx | xxxx | Intent-to-Treat<br>Safety<br>Per-Protocol | xxx<br>xx<br>xx | *********** ******* ****************** |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject and Population (as ordered above).




Date: 24 MAY 2019

## Listing 16.2.4.1: Subject Demographic Information Treatment Group (Page xx of yy)

| Subject | Evaluable | B: Date of Birth<br>A: Age<br>S: Sex | R: Race<br>E: Ethnicity | I: Date of<br>Informed Consent<br>A: Date of Assent | Childbearing<br>Potential | Photography<br>Consent | Protocol<br>Version |
|---|---|---|---|---|---|---|---|
| xxxxx | xxxxxxxx | B: xxxx-xx-xx<br>A: xx<br>S: xxxxxx | R: xxxxxx xxxxxxx<br>xx xxxxx xxxxxxx<br>xxxxxxx | I: xxxx-xx-xx<br>A: xxxx-xx-xx | ХХ | xxx | xxxxxxxxx |
| XXXXX | xxxxxxxx | B: xxxx-xx-xx<br>A: xx<br>S: xxxx | R: xxxxx<br>E: xxxxxxxx xx xxxxxx | I: xxxx-xx-xx<br>A: xxxx-xx-xx | | xxx | xxxxxxxxx |
| XXXXX | xxxxxxxx | B: xxxx-xx-xx<br>A: xx<br>S: xxxxx | R: xxxxx<br>E: xxxxxxx xx xxxxxx | I: xxxx-xx-xx<br>A: xxxx-xx-xx | xxx | xx | xxxxxxxxx |

Note: ITT = Intent-to-Treat Population; S = Safety Population; PP = Per-Protocol Population. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject.




Date: 24 MAY 2019

### Listing 16.2.4.2.1: Unique Medical History Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Medical History Verbatim Term |
|---|---|---|
| XXXX XXX XXXXX | xxxx xxx xxxxx | xxxx |
| | | xxxxxx xxxxxxxxx xx xxxxxx |
| | | xxxxxx xxxxxxxxx xx xxxxx |
| XXXX XXX XXXXX | XXXX XXX XXXXX | XXXX |
| | | xxxxxx xxxxxxxxx xx xxxxxx |
| | | xxxxxx xxxxxxxxx xx xxxxx |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 20.0).
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by System Organ Class, Preferred Term, and Medical History.




Date: 24 MAY 2019

## Listing 16.2.4.2.2: Medical History Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | Condition/Surgery<br>Verbatim Term | P: MedDRA Preferred Term<br>S: MedDRA System Organ Class | S: Start Date (Day) <sup>1</sup> E: End Date (Day) <sup>1</sup> |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxx xxxxxxx xxxxxxxxxx | P: xxxxxx xxxxxxxxx<br>S: xxxxxxxxxxx | S: xxxx-xx-xx (xx)<br>E: xxxxxxx |
| | | | xxxxxxx xxxxxxxx | P: xxxxxxx xxxxxxxx<br>S: xxxxxxxx xxx xxxxxxxx | S: xxxx-xx-xx (xx)<br>E: xxxx-xx-xx (xx) |

Listing sorted by Subject, Medical Condition/Surgery, Start Date, and End Date.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
Note: System Organ Class and Preferred Term map to MedDRA (Version 20.0).
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)




Date: 24 MAY 2019

## Listing 16.2.4.2.3: Substance Use History Treatment Group (Page xx of yy)

| | | | | Alcohol Histor | У | | Smoking Histo | ory | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | Number of Units1 | | | Number | End Date for |
| Subject | Age/Sex | Evaluable | Status | Type of Alcohol <sup>2</sup> | consumed per week | Status | Smoking Type <sup>3</sup> | per day | Ex-Smoker |
| xxxxxx | xxxx | xxxxx | DRINKER | Wine | x | EX-SMOKER | | | xxxx-xx-xx |
| | | | | Beer | х | | | | |
| | | | | Spirits | Х | | | | |
| xxxxxx | xxxx | xxxxxxx | NON-DRINKER | | | NON-SMOKER | | | |
| xxxxx | xxxx | xxxxxxx | NON-DRINKER | | | SMOKER | Cigarettes | X | |
| | | | | | | | E-Cigarettes | Х | |
| | | | | | | | Cigars | X | |
| | | | | | | | Pipes | X | |
| | | | | | | | Smokeless tobacco | X | |
| xxxxx | XXXX | xxxxx | DRINKER | Wine | X | SMOKER | Cigarettes | X | |
| | | | | Beer | X | | E-Cigarettes | Х | |
| | | | | Spirits | X | | Cigars | X | |
| | | | | | | | Pipes | X | |
| | | | | | | | Smokeless tobacco | X | |

<sup>1</sup> Number of units consumed per week (1 unit = 150 mL wine, 360 mL beer, 45 mL spirits)

<sup>&</sup>lt;sup>2</sup> Type of Alcohol is collected on a conditional basis, if "DRINKER", then the number of units consumed per week is collected for each type of alcohol.

<sup>&</sup>lt;sup>3</sup> Smoking Type is collected on a conditional basis, if "SMOKER", then the number of Cigaretts, E-Cigarettes, Cigars, Pipes, and Smokeless tobacco is collected on a per day basis.




Date: 24 MAY 2019

### Listing 16.2.4.4.1: Unique Medication/Therapy Names Coded to WHO-DDE ATC Level 2 Terms and Preferred Names (Page xx of yy)

| ATC Level 2 Term | Preferred Name | Medication/Therapy Name | I: Indication<br>R: Route |
|---|---|---|---|
| xxxxxx xxxxxx xx xxx | xxxxxxxxx | xxxxxxxxx | I: xxxxxxx xxxxxxx<br>R: xxxx |
| | xxxxxxx x | xxxxxx | I: xxxxxxx xxxxxxx<br>xxxxxxxxxxx<br>R: xxxx |
| | xxxxxxxx | xxxxxxxx | I: xxxxxxx xxxxxxx xxxx<br>xxxxx xxxxxxxx<br>R: xxxx |

Note: Preferred Name and ATC Level 2 Term map to the WHO-DDE MAR 2017.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by ATC Level 2 Term, Standardized Medication Name, Medication Name, Indication, and Route.




Date: 24 MAY 2019

## Listing 16.2.4.4.2: Prior and Concomitant Medications/Therapies Treatment Group (Page xx of yy)

| | | | M: Medication/Therapy Name | | D: Dose |
|---|---|---|---|---|---|
| | | | P: Standardized Name | T: Prior/Concomitant | U: Units |
| | | | A: ATC Level 2 Term | S: Start Date/Time (Day) 1 | F: Frequency |
| Subject | Age/Sex | Evaluable | I: Indication | E: End Date/Time (Day) 1 | R: Route |
| xxxxxx | xxxx | xxxxxxxxx | M: xxxxxxxxxxx | T: xxxxxxxxx | D: xx |
| | | | P: xxxxxxxxxxxx | S: xxxx-xx-xxTxx:xx:xx (xx) | U: xx |
| | | | A: xxxxxxxxxxxx | E: xxxx-xx-xxTxx:xx:xx (xx) | F: xxxx |
| | | | I: xxxxxxxx | | R: xxxxxx |
| | | | M: xxxxxxxxxxx | T: xxxxxxxxx | D: xxxxx |
| | | | P: xxxxxxxxxxxx | S: xxxx-xx-xxTxx:xx:xx (xx) | U: xx |
| | | | A: xxxxxxxxxxxx | E: xxxx-xx-xxTxx:xx:xx (xx) | F: xx |
| | | | I: xxxxxxx | | R: xxxx |
| xxxxxx | xxxx | xxxxxxxxx | M: xxxxxxxxxxx | T: xxxxxxxxx | D: xxx |
| | | | P: xxxxxxxxxxxx | S: xxxx-xx-xxTxx:xx:xx (xx) | U: xx |
| | | | A: xxxxxxxxxxxx | E: xxxxxxx | F: xx |
| | | | I: xxxxxxx | | R: xxxx |

Listing sorted by Subject, Start Date, End Date, Medication Name, Indication, and Route. If ongoing, include 'Ongoing' in place of End Date.

¹ Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
Note: Standardized Medication Name and ATC Level 2 Term map to the WHO-DDE (Version MAR 2017).
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)




Date: 24 MAY 2019

### Listing 16.2.4.4.3: Unique Antibiotic Therapy Names Coded to WHO-DDE ATC Level 2 Terms and Preferred Names (Page xx of yy)

| ATC Level 2 Term | Preferred Name | Medication/Therapy Name | I: Indication<br>R: Route |
|---|---|---|---|
| ****** ***** | xxxxxxxxx | xxxxxxxxx | I: xxxxxxx xxxxxxx<br>R: xxxx |
| | xxxxxx x | xxxxxx | I: xxxxxxx xxxxxxx<br>xxxxxxxxxxx<br>R: xxxx |
| | xxxxxxxx | xxxxxxxxx | I: xxxxxxx xxxxxxx xxxx<br>xxxxx xxxxxxx<br>R: xxxx |

Note: Preferred Name and ATC Level 2 Term map to the WHO-DDE MAR 2017.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by ATC Level 2 Term, Standardized Medication Name, Medication Name, Indication, and Route.




Date: 24 MAY 2019

## Listing 16.2.4.4.4: Concomitant Antibiotic Therapies Treatment Group (Page xx of yy)

| | | | M: Medication/Therapy Name | | D: Dose |
|---|---|---|---|---|---|
| | | | P: Standardized Name | T: Prior/Concomitant | U: Units |
| | | | A: ATC Level 2 Term | S: Start Date/Time (Day) 1 | F: Frequency |
| Subject | Age/Sex | Evaluable | I: Indication | E: End Date/Time (Day) 1 | R: Route |
| xxxxx | XXXX | xxxxxxxxx | M: xxxxxxxxxxx | T: xxxxxxxxx | D: xx |
| | | | P: xxxxxxxxxxxx | S: xxxx-xx-xxTxx:xx:xx (xx) | U: xx |
| | | | A: xxxxxxxxxxxx | E: xxxx-xx-xxTxx:xx:xx (xx) | F: xxxx |
| | | | I: xxxxxxx | | R: xxxxxx |
| | | | M: xxxxxxxxxxx | T: xxxxxxxxx | D: xxxxx |
| | | | P: xxxxxxxxxxxx | S: xxxx-xx-xxTxx:xx:xx (xx) | U: xx |
| | | | A: xxxxxxxxxxxx | E: xxxx-xx-xxTxx:xx:xx (xx) | F: xx |
| | | | I: xxxxxxxx | | R: xxxx |
| XXXXXX | xxxx | xxxxxxxxx | M: xxxxxxxxxxx | T: xxxxxxxxx | D: xxx |
| | | | P: xxxxxxxxxxxx | S: xxxx-xx-xxTxx:xx:xx (xx) | U: xx |
| | | | A: xxxxxxxxxxxx | E: xxxxxxx | F: xx |
| | | | I: xxxxxxxx | | R: xxxx |

Listing sorted by Subject, Start Date, End Date, Medication Name, Indication, and Route. If ongoing, include 'Ongoing' in place of End Date.

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
Note: Standardized Medication Name and ATC Level 2 Term map to the WHO-DDE (Version MAR 2017).
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)




Date: 24 MAY 2019

# Listing 16.2.4.6: Physical Examination Treatment Group (Page xx of yy)

| S: Subject A: Age/Sex E: Evaluable | V: Visit<br>D: Date of Exam | H: Height (cm)<br>W: Weight (kg) | Body System Assessed | Result | Abnormal<br>Description | Reason Not Done |
|---|---|---|---|---|---|---|
| S: xxxxx<br>A: xxxx<br>E: xxxxxxxx | V: xxxxxxxxxx<br>D: xxxx-xx-xx | H: xxx<br>W: xx | General Appearance<br>Cardiovascular<br>Neurological<br>Musculoskeletal<br>Extremities/Skin | xxxxxxxx<br>xxxxxxxx<br>xxxxxxxx<br>xxxxxxxx | xxxxxx xxxxxxxx | |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxxx | V: xxxxxxxxxx<br>D: xxxx-xx-xx | H: xxx<br>W: xx | General Appearance<br>Cardiovascular<br>Neurological<br>Musculoskeletal<br>Extremities/Skin | ************************************** | xxxxxxxxxx | ******* ***** **** |
| S: xxxxx<br>A: xxxx<br>E: xxxxxxxx | V: xxxxxxxxxx<br>D: | H:<br>W: | | | | *** *** **** ** |

Listing sorted by Subject, Visit, Date, Body System Assessed.

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)




Date: 24 MAY 2019

# Listing 16.2.5.1: Study Drug Administration Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | Visit | Date/Time<br>of Administration | Where was the<br>Study Drug Administered? | Reason Not Administered |
|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxx | xxxx-xx-xxTxx:xx | xxxxx | |
| | | | XXX XX | xxxx-xx-xxTxx:xx:xx | XXXXXX | |
| | | | XXX XX | xxxx-xx-xxTxx:xx | xxxxx | |
| | | | xxx xx | xxxx-xx-xxTxx:xx:xx | xxxxxx | |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxx | xxxx-xx-xxTxx:xx:xx | xxxxxx | |
| | | | XXX XX | xxxx-xx-xxTxx:xx:xx | XXXXXX | |
| | | | XXX XX | xxxx-xx-xxTxx;xx;xx | xxxxx | |
| | | | XXX XX | | xxx xxxxxxxxx | xx xxxxx xxxxxxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxx | xxxx-xx-xxTxx;xx;xx | xxxxxx | |
| | | | XXX XX | xxxx-xx-xxTxx:xx:xx | xxxxxx | |
| | | | XXX XX | xxxx-xx-xxTxx:xx:xx | xxxxxx | |
| | | | XXX XX | xxxx-xx-xxTxx:xx:xx | XXXXXX | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, visit, Date/Time.




Date: 24 MAY 2019

## Listing 16.2.5.3: Drug Accountability Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | Kit Number | Date<br>Dispensed | Date<br>Returned | Pump ID | Dispensed<br>Weight (units) | Returned<br>Weight (units) |
|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxxx | xxxxx | xxxx-xx-xx | xxxx-xx-xx | Х | xx.xx | xx.xx |
| | | | | | | Х | XX.XX | XX.XX |
| | | | | | | Х | XX.XX | XX.XX |
| | | | | | | Х | xx.xx | XX.XX |
| | | | xxxxx | xxxx-xx-xx | XXXX-XX-XX | Х | xx.xx | XX.XX |
| | | | | | | Х | xx.xx | XX.XX |
| | | | | | | Х | xx.xx | XX.XX |
| | | | | | | X | XX.XX | XX.XX |
| | | | XXXXX | XXXX-XX-XX | XXXX-XX-XX | X | xx.xx | XX.XX |
| | | | | | | X | XX.XX | XX.XX |
| | | | | | | X | XX.XX | XX.XX |
| | | | | | | x | XX.XX | XX.XX |
| xxxxx | xxxx | xxxxxxx | xxxxx | xxxx-xx-xx | xxxx-xx-xx | x | XX.XX | xx.xx |
| | | | | | | X | xx.xx | XX.XX |
| | | | | | | X | xx.xx | XX.XX |
| | | | | | | X | xx.xx | XX.XX |
| | | | XXXXX | XXXX-XX-XX | XXXX-XX-XX | X | xx.xx | XX.XX |
| | | | | | | X | xx.xx | XX.XX |
| | | | | | | X | xx.xx | XX.XX |
| | | | | | | X | XX.XX | XX.XX |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Kit Number, Date Dispensed, Date Returned.




Date: 24 MA

# Listing 16.2.5.4: Dosing Compliance Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex | D: Date of First Dose | Number of<br>Days of | Calculated¹<br>Number of | Amount of<br>Study Drug | Number of | Percent | |
|---|---|---|---|---|---|---|---|
| E: Evaluable | R: Date of Last Dose | Exposure | Doses | Used (g) | Missed Doses | Complaint | Compliant? <sup>2</sup> |
| S: xxxxxx | D: xxxx-xx-xx | xx | xx | xxxx | | xxx | xxx |
| A: xxxx<br>E: xxxxxxxxx | R: xxxx-xx-xx | | | | | | |
| S: xxxxxx | D: xxxx-xx-xx | XX | XX | xxxx | Х | xxx | XX |
| A: xxxx<br>E: xxxxxxxxx | R: xxxx-xx-xx | | | | | | |
| S: xxxxxx | D: xxxx-xx-xx | xx | xx | xxxx | | xxxx | XXX |
| A: xxxx<br>E: xxxxxxxx | R: xxxx-xx-xx | | | | | | |

<sup>1</sup> The total number of doses was calculated from the date of first dose and the date of last known dose minus the missed doses.

 $<sup>^{2}</sup>$  A subject was considered compliant with the dosing regimen if the subject applied at least 80% but no more than 120% of the expected applications.




Date: 24 MAY 2019

## Listing 16.2.5.5: Dosing Deviations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | Date (Day)¹ of<br>Missed Dose | Morning or<br>Afternoon dose? | Reason for Missed Dose |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxx-xx-xx (xx) | xx | ***** |
| | | | xxxx-xx-xx (xx) | xx | XXXXXXX |
| | | | xxxx-xx-xx (xx) | XX | xxxxxx xx |
| xxxxx | xxxx | xxxxxxxx | xxxx-xx-xx (xx) | XX | xxxxxxxx xxxxxxxxx xx xxxxx x xxxxxx |
| | | | xxxx-xx-xx (xx) | xx | XXXXXXXX XXXXXXXXX XX XXXXX X XXXXXXX |
| | | | xxxx-xx-xx (xx) | XX | XXXXXXXX XXXXXXXXXX XX XXXXX X XXXXXXX |
| xxxxx | xxxx | xxxxxxxx | xxxx-xx-xx (xx) | XX | xxxxxx xx |
| | | | xxxx-xx-xx (xx) | xx | XXX XXX |

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)




# Listing 16.2.6.1: Lesion Count Evaluations Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Evaluable | V: Visit D: Date/Time E: Evaluator Initials | Lesion Category | Count | Change<br>from<br>Baseline | Percent Change<br>from Baseline | Reason Not Done |
|---|---|---|---|---|---|---|
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxx | V: SCREENING D: xxxx-xx-xxTxx:xx E: xx | Inflammatory | xx | | | |
| | | Non-Inflammatory | xx | | | |
| | | Total Lesions | XXX | | | |
| | V: BASELINE<br>D: xxxx-xx-xxTxx:xx<br>E: xx | Inflammatory | XX | | | |
| | | Non-Inflammatory | XX | | | |
| | | Total Lesions | XXX | | | |
| | V: DAY 14<br>D: xxxx-xx-xxTxx:xx:xx<br>E: xx | Inflammatory | xx | xx | xxx | |
| | | Non-Inflammatory | XX | x | XXXX | |
| | | Total Lesions | XX | XX | XXXX | |




Listing 16.2.6.2: Investigator Global Assessment
Treatment Group
(Page xx of yy)

Two Grade Reduction from Baseline and S: Subject Two Grade Achieving A: Age/Sex Clear or Evaluator Initials Reduction from E: Evaluable Visit Date/Time Result Baseline Almost Clear or Reason Not Done S: xxxxxx SCREENING xxxx-xx-xxTxx:xx:xx X X XXXXXXX XXX A: xxxx E: xxxxxxxx BASELINE xxxx-xx-xxTxx:xx:xx x x xxxxxxxx XXX DAY 14 xxxx-xx-xxTxx:xx:xx x x xxxxxxxx XX XXXXX DAY 28 xxxx-xx-xxTxx:xx:xx x x xxxxxxxx XX XXX DAY 56 xxxx-xx-xxTxx:xx:xx x x xxxxxxxx XX XX XXX DAY 84 xxxx-xx-xxTxx:xx:xx x x xxxxxxxx XX XXX S: xxxxxx SCREENING xxxx-xx-xxTxx:xx:xx x x xxxxxxxx XXX A: xxxx E: xxxxxxxx BASELINE xxxx-xx-xxTxx:xx:xx x x xxxxxxxx XXX DAY 14 xxxx-xx-xxTxx:xx:xx x x xxxxxxxx XX XX XXX DAY 28 xxxx-xx-xxTxx:xx:xx x x xxxxxxxx XX XX XXX DAY 56 xxxx-xx-xxTxx:xx:xx x x xxxxxxxx XXXX XXX DAY 84 xxxx-xx-xxTxx:xx:xx x x xxxxxxxx XXX

\_\_\_\_\_




Date: 24 MAY 2019

# Listing 16.2.6.3: Patient Reported Outcome Assessment Treatment Group (Page x of xx)

| Subject | Age/Sex | Evaluable | Date of Assessment | Compared to the beginning of treatment, my acne is: | Reason Not Done |
|---|---|---|---|---|---|
| xxxxxxxx | xxxx | xxxxxxxx | xxxx-xx-xx | xxxxx xxxxxxxx | |
| xxxxxxxx | xxxx | xxxxxxxxx | xxxx-xx-xx | xxxxxx xxxxxx | |
| xxxxxxxx | xxxx | xxxxxxxx | xxxx-xx-xx | xxxxx xxxxxxxx | |
| xxxxxxxx | XXXX | xxxxxxxxx | | | xxxxx xxxxxxxx xxxxx |
| xxxxxxxx | XXXX | XXXXXXXXX | xxxx-xx-xx | xxxxx xxxxxxxx | |
| xxxxxxxx | xxxx | xxxxxxxxx | xxxx-xx-xx | xxx xxxxxxx | |




Date: 24 MAY 2019

#### Listing 16.2.6.4: Acne-QoL Questionnaire Treatment Group (Page xx of yy)

| Age/Sex<br>Evaluable | V: Visit<br>D: Date/Time | AQOL Question | Result | Reason<br>Not Done |
|---|---|---|---|---|
| xxxxxx<br>xxx xx<br>xxxxxxx | V: xxxxxxxx<br>D: xxxx-xx-xxTxx:xx:x | х | | xxxxxx xxx<br>xxx xxxx x |
| xxxxxx<br>xxx xx<br>xxxxxxx | V: xxxxxxxx<br>D: xxxx-xx-xxTxx:xx:x | 5. xxxxxxxxx xx xx xxx xxxx xxxx xxx xxx | xxxxx x xxx | |
| | | 6. xx xxx xxxx xxxx xxx xxx xxxxxxxxxx xxx xxx xxxx | xxx xx xxx | |
| | | 8. xx xx xxx xxxx xxxxx xxx xxxxx xxx xx | xxx xx xxx | |
| | | 10. xx xx xxx xxxx xxxx xxx xxxxxxxxxx xxx xxxx | | |
| | | ******* *** *** **** *** *** **** **** **** | xxxxxx x | |
| | | 13. xx xx xxxx xxxx xxxx xxx xxx xxx xxx | XXXXX X | |
| | | 14. xxx xx xxx xxxx xxxxx xxx xxxx xxxx | | |
| | | 15. xxx xx xxx xxxx xxxx xxx xxxxxxx xx xx | | |
| | | 16. xxx xx xxx xxxx xxxxx xxx xxxxxxxx xx | | |
| | | ******** *** *** **** ** *** **** **** **** | | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, AQOL Question.


### Statistical Analysis Plan Botanix BTX.2018.001


Date: 24 MAY 2019

#### Listing 16.2.6.5: Photography Information Treatment Group (Page xx of yy)

| Date of<br>Photograph |
|-----------------------|
| xxxx-xx-xx |
| xxxx-xx-xx |
| xxxx-xx-xx |
| xxxx-xx-xx |
| xxxx-xx-xx |
| xxxx-xx-xx |




Date: 24 MAY 2019

# Listing 16.2.7.1: Cutaneous Tolerability Assessment Treatment Group (Page xx of yy)

| S: Subject | V: Visit | | | | |
|---|---|---|---|---|---|
| | D: Date of assessment | | | Severity | |
| | E: Evaluator Initials | Timepoint | Assessment | Grade <sup>1</sup> | Reason Not Done |
| S: xxxxxx | V: xxxxxxx | Pre-Dose | Burning/Stinging | Х | |
| A: xxxx | D: xxxx-xx-xx | | 3, 3 | | |
| : xxxxxxxx | E: xxx | | | | |
| | | | Dryness | X | |
| | | | Erythema | X | |
| | | | Pruritus | X | |
| | | | Scaling | Х | |
| | | 15 Minutes Post-Dose | Burning/Stinging | х | |
| | | | Dryness | X | |
| | | | Erythema | X | |
| | | | Pruritus | X | |
| | | | Scaling | x | |

Listing sorted by Subject, Visit, Date, Timepoint, Assessment.

<sup>1</sup> Grade 0 = None; Grade 1 = Slight; Grade 2 = Moderate; Grade 3 = Severe.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)




Date: 24 MAY 2019

### Listing 16.2.7.2.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Adverse Event |
|---|---|---|
| xxxx xxx xxxxxxx xxxxxx xxxxxxx | xxxxxxx | xxxxxx |
| | | xxxxxx |
| | xxxxxxxxxx | xxxxxxxxxx |
| xxx xxx xxxxxxxx xxxxxxxx | xxxxxxx | xxxxxxx |
| xxx xxxxxxxx | xxxxxx xxxxxx xxxxxxx | xxxxxxxx xxxxx xxxxxx |
| xxxxxxxxxxxx xxxxxxxx | xxxxxxxx xxxx | xxxxxxxx xxxx |
| | xxxxxxxx xxxxxxxxxx | XXXXX XXXXXXXX XXXXXXXXXX |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 20.0).
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by MedDRA System Organ Class, Preferred Term, and Adverse Event.




Date: 24 MAY 2019

## Listing 16.2.7.2.2: Treatment-Emergent Adverse Events Treatment Group (Page xx of yy)

| : Subject<br>: Age/Sex<br>: Evaluable | A: Adverse Event<br>C: System Organ Class<br>P: Preferred Term | S: Start Date (Day) 1 E: End Date (Day) 1 | S: Severity R: Relationship to Study Drug O: Outcome | S: Is AE Serious? R: Reason(s) for Serious T: Medical Treatment Received? |
|---|---|---|---|---|
| : xxxxxx | A: xxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | G: xxxx | S: xx |
| : xxx xx | C: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: |
| : xxxxxxxx | P: xxxxxxxxxxxxxx | | O: xxxxxxxxx | T: xxx |
| : xxxxxx | A: xxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | G: xxxx | S: xxx |
| : xxx xx | C: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxxxx xxxxxxxx |
| : xxxxxxxxx | P: xxxxxxxxxxxxxx | | O: xxxxxxxxxx | T: xxx |
| : xxxxxx | A: xxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | G: xxxx | S: xxx |
| : xxx xx | C: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxxxxxx xxxxxxxx |
| : xxxxxxxxx | P: xxxxxxxxxxxxxx | | O: xxxxxxxxx | T: xxx |

Programming Notes: If an adverse event is indicated as serious the reason(s) for the event being serious will be listed under the R: Reason(s) for Serious column and serperated by a comma. Possible reason(s) include: Fatal, Life-threatening event, Hospitalization or prolongation of hospitalization, Persistent or significant disability/incapacity, Congenital Anomaly or Birth Defect, Important Medical Event.

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.
Note: System Organ Class and Preferred Term map to MedDRA (Version 20.0).
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)




Date: 24 MAY 2019

## Listing 16.2.7.2.3: Serious Adverse Events Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>A: Evaluable | A: Adverse Event<br>C: System Organ Class<br>P: Preferred Term | S: Start Date (Day) <sup>1</sup> E: End Date (Day) <sup>1</sup> | S: Severity R: Relationship to Study Drug O: Outcome | S: Is AE Serious? R: Reason(s) for Serious T: Medical Treatment Received? |
|---|---|---|---|---|
| S: xxxxxx | A: xxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | G: xxxx | S: xxx |
| : xxx xx | C: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxxxxxxxxx xxxxx xxxxxx |
| : xxxxxxxx | P: xxxxxxxxxxxxxx | | O: xxxxxxxxx | T: xxx |
| : xxxxxx | A: xxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | G: xxxx | S: xxx |
| : xxx xx | C: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxxxx xxxxxxxx |
| : xxxxxxxx | P: xxxxxxxxxxxxxx | | O: xxxxxxxxx | T: xxx |
| : xxxxxx | A: xxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | G: xxxx | S: xxx |
| : xxx xx | C: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxxxxxxx xxxxxxxx |
| : xxxxxxxxx | P: xxxxxxxxxxxxxx | | O: xxxxxxxxx | T: xxx |

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

Note: System Organ Class and Preferred Term map to MedDRA (Version 20.0).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)




Date: 24 MAY 2019

Listing 16.2.7.2.4: Subjects Who Permanently Discontinued Study Drug and/or Discontinued from the Study Due to Adverse Events

Treatment Group

(Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Evaluable | A: Adverse Event<br>C: System Organ Class<br>P: Preferred Term | S: Start Date (Day) <sup>1</sup> E: End Date (Day) <sup>1</sup> | S: Severity R: Relationship to Study Drug O: Outcome | S: Is AE Serious? R: Reason(s) for Serious T: Medical Treatment Received? |
|---|---|---|---|---|
| S: xxxxx<br>A: xxx xx | A: xxxxxxxxxxxxxxxxx<br>C: xxxxxxxxxxxxxxxxx | S: xxxx-xx-xx (xx)<br>E: xxxx-xx-xx (xx) | G: xxxx<br>R: xxxxxxxxx | S: xxx<br>R: xxxxxxxxxxx xxxxx xxxxxx |
| E: xxxxxxxxx | P: xxxxxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | 0: xxxxxxxxx<br>G: xxxx | T: xxx<br>S: xxx |
| A: xxx xx<br>E: xxxxxxxx | C: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | R: xxxxxxxxx<br>O: xxxxxxxxx | R: xxxxxx xxxxxxxx<br>T: xxx |
| S: xxxxxx<br>A: xxx xx<br>E: xxxxxxxx | A: xxxxxxxxxxxxxxxx<br>C: xxxxxxxxxxxxxxx<br>P: xxxxxxxxxxxxxxxxx | S: xxxx-xx-xx (xx)<br>E: xxxx-xx-xx (xx) | G: xxxx<br>R: xxxxxxxxx<br>O: xxxxxxxxx | S: xxx<br>R: xxxxxxxxx xxxxxxxx<br>T: xxx |

<sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
 date - date of first dose + 1 for dates on or after first dose.
Note: System Organ Class and Preferred Term map to MedDRA (Version 20.0).
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)




Date: 24 MAY 2019

Listing 16.2.7.2.5: Unique Abuse-Related Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Adverse Event |
|---|---|---|
| XXXXX XXX XXXXXXXX XXXXXXX | xxxxxxx | xxxxxx |
| | | xxxxxx |
| | xxxxxxxxxx | xxxxxxxxxx |
| xxx xxx xxxxxxxx xxxxxxxx | xxxxxxx | xxxxxxx |
| xxx xxxxxxxx | xxxxxx xxxxxx xxxxxxx | xxxxxxxx xxxxx xxxxx |
| xxxxxxxxxxxx xxxxxxxx | xxxxxxxx xxxx | xxxxxxxx xxxx |
| | xxxxxxxx xxxxxxxxxx | xxxxx xxxxxxxx xxxxxxxxxx |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 20.0). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by MedDRA System Organ Class, Preferred Term, and Adverse Event.




Date: 24 MAY 2019

## Listing 16.2.7.2.6: Treatment-Emergent Abuse-Related Adverse Events Treatment Group (Page xx of yy)

| : Subject<br>: Age/Sex<br>: Evaluable | A: Adverse Event<br>C: System Organ Class<br>P: Preferred Term | S: Start Date (Day) <sup>1</sup> E: End Date (Day) <sup>1</sup> | S: Severity R: Relationship to Study Drug O: Outcome | S: Is AE Serious? R: Reason(s) for Serious T: Medical Treatment Received? |
|---|---|---|---|---|
| : xxxxxx | A: xxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | G: xxxx | S: xx |
| : xxx xx | C: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: |
| : xxxxxxxx | P: xxxxxxxxxxxxxx | | O: xxxxxxxxx | T: xxx |
| : xxxxxx | A: xxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | G: xxxx | S: xxx |
| : xxx xx | C: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxxxx xxxxxxxx |
| : xxxxxxxxx | P: xxxxxxxxxxxxxx | | O: xxxxxxxxx | T: xxx |
| : xxxxxx | A: xxxxxxxxxxxxx | S: xxxx-xx-xx (xx) | G: xxxx | S: xxx |
| : xxx xx | C: xxxxxxxxxxxxxx | E: xxxx-xx-xx (xx) | R: xxxxxxxxxx | R: xxxxxxxx xxxxxxxx |
| : xxxxxxxxx | P: xxxxxxxxxxxxxx | | O: xxxxxxxxx | T: xxx |

Programming Notes: If an adverse event is indicated as serious the reason(s) for the event being serious will be listed under the R: Reason(s) for Serious column and serperated by a comma. Possible reason(s) include: Fatal, Life-threatening event, Hospitalization or prolongation of hospitalization, Persistent or significant disability/incapacity, Congenital Anomaly or Birth Defect, Important Medical Event.

Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as
date - date of first dose + 1 for dates on or after first dose.

Note: System Organ Class and Preferred Term map to MedDRA (Version 20.0).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)




Date: 24 MAY 2019

# Listing 16.2.8.1: Urine Pregnancy Test Results Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | Visit | Date/Time | Results |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxx-xx-xxTxx:xx | xxxxxxx |
| | | | xxxxxxxx | xxxx-xx-xxTxx:xx | xxxxxxxx |
| | | | xxx xx | xxxx-xx-xxTxx:xx:xx | xxxxxxxx |
| | | | xxx xx | xxxx-xx-xxTxx:xx:xx | xxxxxxx |
| | | | XXX XX | xxxx-xx-xxTxx:xx:xx | xxxxxxx |
| XXXXX | XXXX | xxxxxxxx | xxxxxxxx | xxxx-xx-xxTxx:xx | xxxxxxx |
| | | | xxxxxxx | xxxx-xx-xxTxx:xx:xx | XXXXXXX |
| | | | XXX XX | xxxx-xx-xxTxx:xx:xx | XXXXXXX |
| | | | XXXX XXXXXXXX | xxxx-xx-xxTxx:xx | xxxxxxx |
| XXXXX | XXXX | xxxxxxxx | xxxxxxxx | xxxx-xx-xxTxx:xx | xxxxxxx |
| | | | xxxxxxx | xxxx-xx-xxTxx:xx | xxxxxxx |
| | | | xxx xx | xxxx-xx-xxTxx;xx;xx | xxxxxxx |
| | | | xxx xx | xxxx-xx-xxTxx:xx | xxxxxxx |
| | | | xxxx xxxxxxxx | xxxx-xx-xxTxx:xx | XXXXXXX |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Date.




Date: 24 MAY 2019

## Listing 16.2.8.2: Urine Drug Screen Results Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | Visit | Date/Time | Results | Positive Drugs | Reason Not Done |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxx-xx-xxTxx;xx<br>xxxx-xx-xxTxx;xx | xxxxxxx | xxxxxxxxx | |
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx<br>xxxxxxxx | xxxx-xx-xxTxx:xx | xxxxxxx | | xxxxx xxxxxxx |
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxx-xx-xxTxx:xx<br>xxxx-xx-xxTxx:xx | xxxxxxx | ************************************** | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Programming Notes: The Positive Drugs column will list all of the drugs that apply as positive or (Yes) for the drug screen, each separated by a comma. For example if the Result is Positive and the drug screen found Amphetamines and Methamphetamines as Positive then they will be listed as Amphetamines, Methamphetamines.

Listing sorted by Subject, Visit, Date.




Listing 16.2.8.2.1.1: Complete Blood Count Laboratory Test Results

Treatment Group

(Page xx of yy)

\_\_\_\_\_

| A: Age/Sex | V: Visit | | Results | | Referenc | e Range | Reason Not Done/ |
|---|---|---|---|---|---|---|---|
| E: Evaluable | D: Date/Time | Laboratory Test | (Units) | Low | High | Indicator (CS1) | Comments |
| 3: xxxxx<br>A: xxxx<br>E: xxxxxxxx | V: xxxxxxxxx<br>D: xxxx-xx-xxTxx:xx | ****** | xxx xxx | х | XX | ***** | |
| | | xxxxxxxxxx | XXX XXXXXX | xx | XX | xxxxxx xxxx | |
| | | xxxxxxxxxxxxx | XXX XXXXXX | xx | XX | xxxxxx xxxx | |
| | | xxxxxxxxxxxxx | xxx xxxxxx | XX | XX | xxxxxx xxxx | |
| | V: xxxxxxxx<br>D: xxxx-xx-xxTxx:xx:xx | xxxxxxx | xxx xxxxxx | XX | xx | xxxxxx xxxx | |
| | | xxxxxxxxxxxx | XXX XXXXXX | XX | XX | xxxxxx xxxx | |
| | | xxxxxxxxxxxxxxx | XXX XXXXXX | XX | XX | xxxxxx xxxx | |
| | | xxxxxxxxxxxxxxx | | | | | xxx xxx xxxxx |
| | | | | | | | xxxxxxxxxx xxxx |
| | V: xxxxxxxx<br>D: xxxx-xx-xxTxx:xx:xx | xxxxxxxxxxxxxx | xxx xxxxxx | XX | xx | xxxxxx xxxxx | |
| | | xxxxxx xxxxxxx | XXX XXXXXX | XX | XX | xxxxxx xxxx | |
| | | xxxxxxxxxx | XXX XXX | X | XX | xxxxxx xxxx | |
| | | xxxxxxxxxxxxxxxx | XXX XXX | Х | XX | xxxxxx xxxx | |

Listing sorted by Subject, Visit, Date/Time, and Lab Test.

<sup>1</sup> Clinically Significant per Investigator SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)




Date: 24 MAY 2019

Repeat Listing 16.2.8.2.1.1: for the following listings: Listing 16.2.8.2.1.2: Chemistry Laboratory Test Results

Listing 16.2.8.2.1.3: Urinalysis Laboratory Test Results